CLINICAL TRIAL: NCT03197376
Title: A Phase 3, Randomized, Double-Blind Study of the Safety, Tolerability, Lot-to-Lot Consistency, Immunogenicity & Non-Interference With Concomitant Vaccinations of Serum Institute of PNEUMOSIL in Healthy Infants in The Gambia
Brief Title: Phase 3 Study of 10-valent Pneumococcal Conjugate Vaccine (PNEUMOSIL) in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAC-056
Record Dates: First submitted 2017-06-21; First posted 2017-06-23 (Actual); Results first posted 2019-09-11 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2019-08

CONDITIONS: Pneumonia, Pneumococcal
MeSH Terms: conditions — Pneumonia, Pneumococcal | interventions — PHiD-CV vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pneumosil Lot 1 (Experimental): Pneumosil Lot 1
  Interventions: Biological: Pneumosil
- Pneumosil Lot 2 (Experimental): Pneumosil Lot 2
  Interventions: Biological: Pneumosil
- Pneumosil Lot 3 (Experimental): Pneumosil Lot 3
  Interventions: Biological: Pneumosil
- Synflorix (Active Comparator): Synflorix
  Interventions: Biological: Synflorix

INTERVENTIONS:
Biological: Pneumosil — 10-Valent Pneumococcal Conjugate Vaccine
  Arms: Pneumosil Lot 1; Pneumosil Lot 2; Pneumosil Lot 3
Biological: Synflorix — Pneumococcal conjugate vaccine (Non-Typeable Haemophilus influenzae (NTHi) protein D, diphtheria or tetanus toxoid conjugates) adsorbed
  Arms: Synflorix

SUMMARY:
This study will examine the consistency of 3 batches of the Pneumosil vaccine by looking at the immune response in infants. In addition, the study will compare the immunogenicity of the Pneumosil vaccine to another WHO-prequalified vaccine, Synflorix.

DETAILED DESCRIPTION:
This is a randomized, active-controlled, double-blind, Phase 3 study in 2,250 healthy infants (6 to 8 weeks of age). Subjects will receive 3 doses of either PNEUMOSIL (3 groups receiving vaccine from different lots) or Synflorix (1 group) at 6, 10, and 14 weeks of age. The first 675 randomized subjects will receive a booster dose of either PNEUMOSIL or Synflorix at 9 months of age that matches the treatment assignment for the priming phase. Standard EPI vaccinations in The Gambia will be given concomitantly with all 4 doses of the study vaccines. Out of the 675 booster subjects, subjects who consented for further evaluation will participate for the assessment of immune persistence 12 (+1) months after the booster vaccination

The primary objectives are to demonstrate that the three lots of the Pneumosil vaccine is consistent by evaluating the immune responses, and to demonstrate that the immune responses generated by Pneumosil are non-inferior to those generated by Synflorix. The safety and tolerability of Pneumosil will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* They are healthy infants based on medical history and clinical assessment.
* They are between 6 and 8 weeks (ie 42 to 56 days) old, inclusive.
* Subject's parent must provide voluntary written/thumb-printed informed consent and be willing to comply with study requirements and procedures.

Exclusion Criteria:

* Use of any investigational medicinal product prior to randomization.
* Previous vaccination against or infection with S. pneumoniae.
* History of anaphylactic shock or an allergic reaction to any prior vaccination.
* Any fever, illness (including malaria).
* Receipt of another vaccine within 30 days of study start.
* Chronic administration of an immunosuppressant or administration of immunoglobulins
* History of blood disorder, primary immunodeficiency, or a sibling who has such a diagnosis or who died of suddenly without apparent cause.
* History of meningitis, seizures or any neurological disorder.

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2250 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2019-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ed Clarke, Principal Investigator — Medical Research Council (MRC) Unit, The Gambia
Locations (1):
- Medical Research Council (MRC) Unit, The Gambia, Fajara, The Gambia

REFERENCES:
- [Derived] Clarke E, Bashorun A, Adigweme I, Badjie Hydara M, Umesi A, Futa A, Ochoge M, Obayemi D, Edem B, Saidy-Jah E, Onwuchekwa C, Dhere R, Sethna V, Kampmann B, Goldblatt D, Taylor D, Andi-Lolo I, Hosken N, Antony K, Innis BL, Alderson MR, Lamola S. Immunogenicity and safety of a novel ten-valent pneumococcal conjugate vaccine in healthy infants in The Gambia: a phase 3, randomised, double-blind, non-inferiority trial. Lancet Infect Dis. 2021 Jun;21(6):834-846. doi: 10.1016/S1473-3099(20)30735-0. Epub 2021 Jan 28. PMID 33516293

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 21 June 2017 to 29 January 2018
Pre-assignment Details: Randomization took place only after a subject had satisfied all eligibility criteria. Subjects were randomized in a 2:2:2:3 ratio based on a pre-established randomization scheme.
Groups:
- Pneumosil Lot 1: 10-Valent Pneumococcal Conjugate Vaccine Lot 1
- Pneumosil Lot 2: 10-Valent Pneumococcal Conjugate Vaccine Lot 2
- Pneumosil Lot 3: 10-Valent Pneumococcal Conjugate Vaccine Lot 3
Period: Primary and Booster Phase
Arm/Group | Pneumosil Lot 1 | Pneumosil Lot 2 | Pneumosil Lot 3 | Synflorix
Started | 502 | 501 | 500 | 747
Vaccinated-Dose 1 | 502 | 501 | 500 | 747
Vaccinated-Dose 2 | 495 | 495 | 491 | 738
Vaccinated-Dose 3 | 492 | 493 | 490 | 731
Primary Reactogenicity Cohort | 251 | 243 | 257 | 364
Booster Cohort | 150 | 151 | 150 | 224
Received Booster Vaccine | 145 | 144 | 139 | 213
Completed (Completed main phase of study excluding immune persistence phase) | 487 | 488 | 480 | 722
Not Completed | 15 | 13 | 20 | 25
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Death | 1 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 1 | 3
Not completed — Withdrawal by subject's parents | 11 | 10 | 14 | 11
Not completed — Ineligibility criteria | 1 | 1 | 4 | 2
Not completed — Not vaccine related | 1 | 2 | 0 | 6
Period: Immune Persistence Phase
Arm/Group | Pneumosil Lot 1 | Pneumosil Lot 2 | Pneumosil Lot 3 | Synflorix
Started | 132 | 133 | 128 | 195
Completed | 127 | 129 | 123 | 190
Not Completed | 5 | 4 | 5 | 5
Not completed — Lost to Follow-up | 0 | 0 | 2 | 1
Not completed — Withdrawal by subject's parents | 4 | 4 | 2 | 3
Not completed — Not vaccine related | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Pneumosil Lot 1: Three doses of Pneumosil Lot 1
- Pneumosil Lot 2: Three doses of Pneumosil Lot 2
- Pneumosil Lot 3: Three doses of Pneumosil Lot 3
- Synflorix: Three doses of Synflorix
- Total: Total of all reporting groups
Arm/Group | Pneumosil Lot 1 | Pneumosil Lot 2 | Pneumosil Lot 3 | Synflorix | Total
Number analyzed (Participants) | 502 | 501 | 500 | 747 | 2250
Age, Continuous [Mean (Standard Deviation); unit: Days] — Age at enrollment in days
  Days | 47.0 (3.78) | 47.1 (4.10) | 47.3 (4.03) | 47.1 (4.05) | 47.2 (4.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 252 | 241 | 245 | 347 | 1085
  Male | 250 | 260 | 255 | 400 | 1165
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race-African | 502 | 500 | 500 | 747 | 2249
  Race-Other | 0 | 1 | 0 | 0 | 1
  Ethnicity-Mandinka | 264 | 256 | 257 | 397 | 1174
  Ethnicity-Wolof | 47 | 58 | 51 | 61 | 217
  Ethnicity-Fula | 61 | 63 | 62 | 86 | 272
  Ethnicity-Jola | 63 | 54 | 63 | 100 | 280
  Ethnicity-Serahule | 11 | 16 | 20 | 29 | 76
  Ethnicity-Serere | 21 | 14 | 13 | 21 | 69
  Ethnicity-Manjago | 8 | 11 | 5 | 11 | 35
  Ethnicity-Other | 26 | 29 | 29 | 42 | 126
Region of Enrollment [Number; unit: participants]
  Gambia | 502 | 501 | 500 | 747 | 2250

OUTCOME MEASURES:

1. Primary Outcome: Serotype-specific Geometric Mean Concentration of IgG Antibody
Description: Serotype-specific concentrations of immunoglobulin G (IgG) antibody measured by ELISA
Time Frame: 4 weeks after the third dose
Population: All subjects who received all primary series doses of study vaccines, had post-dose immunogenicity measurement(s) with no major protocol deviations
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Groups:
- Lot 1: Three doses of Pneumosil Lot 1
- Lot 2: Three doses of Pneumosil Lot 2
- Lot 3: Three doses of Pneumosil Lot 3
Arm/Group | Lot 1 | Lot 2 | Lot 3
Number analyzed (Participants) | 487 | 490 | 481
µg/mL
  Pn IgG Type 1 | 4.08 [3.84 to 4.33] | 4.24 [3.97 to 4.52] | 4.58 [4.30 to 4.87]
  Pn IgG Type 5 | 1.34 [1.27 to 1.43] | 1.80 [1.70 to 1.91] | 1.84 [1.73 to 1.96]
  Pn IgG Type 6A | 1.05 [0.95 to 1.15] | 0.95 [0.86 to 1.06] | 1.01 [0.91 to 1.11]
  Pn IgG Type 6B: number analyzed (Participants) | 484 | 488 | 480
  Pn IgG Type 6B | 1.30 [1.15 to 1.47] | 0.92 [0.81 to 1.05] | 1.49 [1.32 to 1.68]
  Pn IgG Type 7F | 2.79 [2.61 to 2.98] | 2.55 [2.37 to 2.75] | 3.70 [3.46 to 3.96]
  Pn IgG Type 9V | 1.28 [1.20 to 1.37] | 1.19 [1.11 to 1.28] | 1.46 [1.36 to 1.56]
  Pn IgG Type 14: number analyzed (Participants) | 487 | 489 | 480
  Pn IgG Type 14 | 4.99 [4.52 to 5.51] | 5.37 [4.87 to 5.92] | 5.25 [4.78 to 5.76]
  Pn IgG Type 19A: number analyzed (Participants) | 483 | 490 | 481
  Pn IgG Type 19A | 1.53 [1.42 to 1.66] | 1.66 [1.53 to 1.79] | 1.74 [1.61 to 1.88]
  Pn IgG Type 19F: number analyzed (Participants) | 484 | 489 | 480
  Pn IgG Type 19F | 4.20 [3.92 to 4.50] | 5.02 [4.68 to 5.39] | 3.89 [3.59 to 4.21]
  Pn IgG Type 23F: number analyzed (Participants) | 487 | 489 | 481
  Pn IgG Type 23F | 1.61 [1.48 to 1.74] | 1.57 [1.44 to 1.72] | 1.56 [1.44 to 1.70]
Statistical Analysis 1: Comparison: Lot 1 vs Lot 2; The 3 lots were to be considered equivalent if, for each serotype, all 3 CIs for IgG GMC ratios 4 weeks after the primary vaccination series lay within the interval (0.5, 2); Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for each serotype 1, Lot 1 and Lot 2 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 1 GMC Ratio = 0.96, 95% CI 2-sided [0.88 to 1.05]
Statistical Analysis 2: Comparison: Lot 1 vs Lot 2; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 5, Lot 1 and Lot 2 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 5 GMC Ratio = 0.75, 95% CI 2-sided [0.69 to 0.81]
Statistical Analysis 3: Comparison: Lot 1 vs Lot 2; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 6A, Lot 1 and Lot 2 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 6A GMC Ratio = 1.1, 95% CI 2-sided [0.96 to 1.26]
Statistical Analysis 4: Comparison: Lot 1 vs Lot 2; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 6B, Lot 1 and Lot 2 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 6B GMC Ratio = 1.41, 95% CI 2-sided [1.18 to 1.69]
Statistical Analysis 5: Comparison: Lot 1 vs Lot 2; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 7F, Lot 1 and Lot 2 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 7F GMC Ratio = 1.09, 95% CI 2-sided [0.99 to 1.20]
Statistical Analysis 6: Comparison: Lot 1 vs Lot 2; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 9V, Lot 1 and Lot 2 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 9V GMC Ratio = 1.08, 95% CI 2-sided [0.98 to 1.18]
Statistical Analysis 7: Comparison: Lot 1 vs Lot 2; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 14, Lot 1 and Lot 2 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 14 GMC Ratio = 0.93, 95% CI 2-sided [0.81 to 1.07]
Statistical Analysis 8: Comparison: Lot 1 vs Lot 2; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 19A, Lot 1 and Lot 2 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 19A GMC Ratio = 0.93, 95% CI 2-sided [0.83 to 1.04]
Statistical Analysis 9: Comparison: Lot 1 vs Lot 2; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 19F, Lot 1 and Lot 2 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 19F GMC Ratio = 0.84, 95% CI 2-sided [0.76 to 0.92]
Statistical Analysis 10: Comparison: Lot 1 vs Lot 2; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 23F, Lot 1 and Lot 2 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 23F GMC Ratio = 1.02, 95% CI 2-sided [0.91 to 1.15]
Statistical Analysis 11: Comparison: Lot 1 vs Lot 3; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 1, Lot 1 and Lot 3 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 1 GMC Ratio = 0.89, 95% CI 2-sided [0.82 to 0.97]
Statistical Analysis 12: Comparison: Lot 1 vs Lot 3; The 3 lots were to be considered equivalent if, for each serotype, all 3 CIs for IgG GMC ratios 4 weeks after the primary vaccination series lay within the interval (0.5, 2; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 5, Lot 1 and Lot 3 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 5 GMC Ratio = 0.73, 95% CI 2-sided [0.67 to 0.80]
Statistical Analysis 13: Comparison: Lot 1 vs Lot 3; [analysis description as in outcome 1, analysis 12]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 6A, Lot 1 and Lot 3 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 6A GMC Ratio = 1.04, 95% CI 2-sided [0.91 to 1.20]
Statistical Analysis 14: Comparison: Lot 1 vs Lot 3; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 6B, Lot 1 and Lot 3 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 6B GMC Ratio = 0.87, 95% CI 2-sided [0.74 to 1.04]
Statistical Analysis 15: Comparison: Lot 1 vs Lot 3; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 7F, Lot 1 and Lot 3 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 7F GMC Ratio = 0.75, 95% CI 2-sided [0.68 to 0.83]
Statistical Analysis 16: Comparison: Lot 1 vs Lot 3; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 9V, Lot 1 and Lot 3 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 9V GMC Ratio = 0.88, 95% CI 2-sided [0.80 to 0.97]
Statistical Analysis 17: Comparison: Lot 1 vs Lot 3; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 14, Lot 1 and Lot 3 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 14 GMC Ratio = 0.95, 95% CI 2-sided [0.83 to 1.09]
Statistical Analysis 18: Comparison: Lot 1 vs Lot 3; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 19A, Lot 1 and Lot 3 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 19A GMC Ratio = 0.88, 95% CI 2-sided [0.79 to 0.98]
Statistical Analysis 19: Comparison: Lot 1 vs Lot 3; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 19F, Lot 1 and Lot 3 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 19F GMC Ratio = 1.08, 95% CI 2-sided [0.97 to 1.20]
Statistical Analysis 20: Comparison: Lot 1 vs Lot 3; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 24F, Lot 1 and Lot 3 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 23F GMC Ratio = 1.03, 95% CI 2-sided [0.92 to 1.15]
Statistical Analysis 21: Comparison: Lot 2 vs Lot 3; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 1, Lot 2 and Lot 3 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 1 GMC Ratio = 0.93, 95% CI 2-sided [0.85 to 1.01]
Statistical Analysis 22: Comparison: Lot 2 vs Lot 3; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 5, Lot 2 and Lot 3 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 5 GMC Ratio = 0.98, 95% CI 2-sided [0.90 to 1.07]
Statistical Analysis 23: Comparison: Lot 2 vs Lot 3; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 6A, Lot 2 and Lot 3 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 6A GMC Ratio = 0.95, 95% CI 2-sided [0.82 to 1.09]
Statistical Analysis 24: Comparison: Lot 2 vs Lot 3; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 6B, Lot 2 and Lot 3 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 6B GMC Ratio = 0.62, 95% CI 2-sided [0.52 to 0.74]
Statistical Analysis 25: Comparison: Lot 2 vs Lot 3; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 7F, Lot 2 and Lot 3 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 7F GMC Ratio = 0.69, 95% CI 2-sided [0.62 to 0.76]
Statistical Analysis 26: Comparison: Lot 2 vs Lot 3; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 9V, Lot 2 and Lot 3 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 9V GMC Ratio = 0.82, 95% CI 2-sided [0.74 to 0.90]
Statistical Analysis 27: Comparison: Lot 2 vs Lot 3; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 14, Lot 2 and Lot 3 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 14 GMC Ratio = 1.02, 95% CI 2-sided [0.89 to 1.17]
Statistical Analysis 28: Comparison: Lot 2 vs Lot 3; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 19A, Lot 2 and Lot 3 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 19A GMC Ratio = 0.95, 95% CI 2-sided [0.85 to 1.06]
Statistical Analysis 29: Comparison: Lot 2 vs Lot 3; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 19F, Lot 2 and Lot 3 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 19F GMC Ratio = 1.29, 95% CI 2-sided [1.16 to 1.44]
Statistical Analysis 30: Comparison: Lot 2 vs Lot 3; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the GMC of IgG antibody at one month following third vaccination was within this equivalence interval for serotype 23F, Lot 2 and Lot 3 would be equivalent with respect to the immune response to the vaccine lot; Pn IgG type 23F GMC Ratio = 1.00, 95% CI 2-sided [0.89 to 1.13]

2. Primary Outcome: Number and Percentage of Subjects With Serotype-specific IgG Antibody Responses ≥ 0.35 μg/mL
Description: Number and Percentage of subjects with serotype-specific IgG Antibody Responses ≥ 0.35 μg/mL
Time Frame: 4 weeks after the third dose
Population: Non-inferiority for each serotype is based on 2 non-inferiority criteria evaluation: for each serotype, non-inferiority was shown if a two-sided 97.5% CI for the absolute difference in proportions responding (PNEUMOSIL-Synflorix) had a lower limit >-0.10, or if a two-sided 97.5% CI for the IgG GMC ratio (PNEUMOSIL/Synflorix) had a lower limit >0.5.
Measure: Count of Participants; unit: Participants
Groups:
- Pneumosil: Three doses of Pneumosil
Arm/Group | Pneumosil | Synflorix
Number analyzed (Participants) | 1458 | 724
Participants
  Pn IgG Type 1 | 1454 | 717
  Pn IgG Type 5 | 1435 | 692
  Pn IgG Type 6A | 1193 | 555
  Pn IgG Type 6B: number analyzed (Participants) | 1452 | 724
  Pn IgG Type 6B | 1142 | 555
  Pn IgG Type 7F | 1443 | 709
  Pn IgG Type 9V | 1391 | 690
  Pn IgG Type 14: number analyzed (Participants) | 1456 | 722
  Pn IgG Type 14 | 1437 | 715
  Pn IgG Type 19A: number analyzed (Participants) | 1454 | 724
  Pn IgG Type 19A | 1386 | 555
  Pn IgG Type 19F: number analyzed (Participants) | 1453 | 720
  Pn IgG Type 19F | 1427 | 713
  Pn IgG Type 23F: number analyzed (Participants) | 1457 | 724
  Pn IgG Type 23F | 1372 | 557
Statistical Analysis 1: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — Non-inferiority was to be shown if either the lower limit of the 97.5% CI for the difference in proportions of IgG responders (PNEUMOSIL-Synflorix) exceeded -10%, for 7 or more of the 10 serotypes in PNEUMOSIL; Absolute Difference for Type 1 = 0.7, 97.5% CI 2-sided [-0.0 to 1.9]
Statistical Analysis 2: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — Non-inferiority was to be shown if either the lower limit of the 97.5% CI for the difference in proportions of IgG responders (PNEUMOSIL-Synflorix) exceeded -10% for 7 or more of the 10 serotypes in PNEUMOSIL; Absolute Difference for Type 5 = 2.8, 97.5% CI 2-sided [1.2 to 5.0]
Statistical Analysis 3: Comparison: Pneumosil vs Synflorix; Synflorix proportion of responders for serotype 6A was operationally defined as the lowest observed proportion of responders among the 8 serotypes in common with PNEUMOSIL; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 2]; Absolute Difference for Type 6A = 5.2, 97.5% CI 2-sided [1.1 to 9.5]
Statistical Analysis 4: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 2]; Absolute Difference for Type 6B = 2.0, 97.5% CI 2-sided [-2.2 to 6.4]
Statistical Analysis 5: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 2]; Absolute Difference for Type 7F = 1.0, 97.5% CI 2-sided [-0.1 to 2.7]
Statistical Analysis 6: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 2]; Absolute Difference for Type 9V = 0.1, 97.5% CI 2-sided [-1.9 to 2.5]
Statistical Analysis 7: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 2]; Absolute Difference for Type 14 = -0.3, 97.5% CI 2-sided [-1.4 to 1.0]
Statistical Analysis 8: Comparison: Pneumosil vs Synflorix; Synflorix proportion of responders for serotype 19A was operationally defined as the lowest observed proportion of responders among the 8 serotypes in common with PNEUMOSIL; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 2]; Absolute Difference for Type 19A = 18.7, 97.5% CI 2-sided [15.1 to 22.5]
Statistical Analysis 9: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 2]; Absolute Difference for Type 19F = -0.8, 97.5% CI 2-sided [-1.9 to 0.5]
Statistical Analysis 10: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 2]; Absolute Difference for Type 23F = 17.2, 97.5% CI 2-sided [13.6 to 21.1]

3. Primary Outcome: Serotype-specific Geometric Mean Concentration of IgG Antibody
Description: Serotype-specific immunoglobulin G (IgG) geometric mean concentration (GMC) 4 weeks after the primary series of PNEUMOSIL/Synflorix co-administered with pentavalent, RV and polio vaccines.
Time Frame: 4 weeks after the third dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Groups:
- Pneumosil: IgG GMC after three doses of Pneumosil
- Synflorix: IgG GMC after three doses of Synflorix
Arm/Group | Pneumosil | Synflorix
Number analyzed (Participants) | 1458 | 724
µg/mL
  Pn IgG Type 1 | 4.29 [4.14 to 4.45] | 1.99 [1.88 to 2.11]
  Pn IgG Type 5 | 1.65 [1.59 to 1.71] | 1.20 [1.14 to 1.26]
  Pn IgG Type 6A | 1.00 [0.95 to 1.06] | 1.13 [1.02 to 1.25]
  Pn IgG Type 6B: number analyzed (Participants) | 1452 | 724
  Pn IgG Type 6B | 1.21 [1.13 to 1.30] | 1.13 [1.02 to 1.25]
  Pn IgG Type 7F | 2.97 [2.85 to 3.10] | 2.29 [2.16 to 2.43]
  Pn IgG Type 9V | 1.31 [1.26 to 1.36] | 1.42 [1.34 to 1.50]
  Pn IgG Type 14: number analyzed (Participants) | 1456 | 722
  Pn IgG Type 14 | 5.20 [4.92 to 5.50] | 4.24 [3.90 to 4.61]
  Pn IgG Type 19A: number analyzed (Participants) | 1454 | 724
  Pn IgG Type 19A | 1.64 [1.57 to 1.72] | 1.13 [1.02 to 1.25]
  Pn IgG Type 19F: number analyzed (Participants) | 1453 | 720
  Pn IgG Type 19F | 4.35 [4.17 to 4.54] | 5.93 [5.50 to 6.39]
  Pn IgG Type 23F: number analyzed (Participants) | 1457 | 724
  Pn IgG Type 23F | 1.58 [1.51 to 1.66] | 0.87 [0.80 to 0.95]
Statistical Analysis 1: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — Non-inferiority was to be shown if the lower limit of the 97.5% CI for the GMC ratio (PNEUMOSIL/Synflorix) exceeded 0.5, for 7 or more of the 10 serotypes in PNEUMOSIL; Pn IgG type 1 GMC Ratio = 2.15, 97.5% CI 2-sided [2.00 to 2.32]
Statistical Analysis 2: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Pn IgG type 5 GMC Ratio = 1.37, 97.5% CI 2-sided [1.28 to 1.47]
Statistical Analysis 3: Comparison: Pneumosil vs Synflorix; [analysis description as in outcome 2, analysis 3]; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Pn IgG type 6A GMC Ratio = 0.89, 97.5% CI 2-sided [0.78 to 1.01]
Statistical Analysis 4: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Pn IgG type 6B GMC Ratio = 1.07, 97.5% CI 2-sided [0.93 to 1.24]
Statistical Analysis 5: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Pn IgG type 7F GMC Ratio = 1.30, 97.5% CI 2-sided [1.19 to 1.41]
Statistical Analysis 6: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Pn IgG type 9V GMC Ratio = 0.92, 97.5% CI 2-sided [0.85 to 1.00]
Statistical Analysis 7: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Pn IgG type 14 GMC Ratio = 1.23, 97.5% CI 2-sided [1.10 to 1.37]
Statistical Analysis 8: Comparison: Pneumosil vs Synflorix; [analysis description as in outcome 2, analysis 8]; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Pn IgG type 19A GMC Ratio = 1.45, 97.5% CI 2-sided [1.30 to 1.63]
Statistical Analysis 9: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Pn IgG type 19F GMC Ratio = 0.73, 97.5% CI 2-sided [0.67 to 0.80]
Statistical Analysis 10: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Pn IgG type 23F GMC Ratio = 1.81, 97.5% CI 2-sided [1.63 to 2.01]

4. Primary Outcome: Number and Percentage of Subjects With EPI Vaccine Immune Responses (Diphtheria, Tetanus, Hepatitis B, Hib, Polio and Rotavirus)
Description: Subjects with 1) anti-diphtheria toxoid (DT) and anti-tetanus toxoid (DT) IgG concentration ≥ 0.1 IU/mL; 2) anti-Hepatitis B surface antigen (HBsAg) IgG concentration ≥ 10 mIU/mL; 3) anti-Hib (polyribosylribitol phosphate [PRP]) IgG concentration ≥ 0.15 µg/mL; 4) anti-poliovirus types 1, 2 and 3 neutralizing antibody titers ≥ 1:8; 5) anti-rotavirus IgA concentration ≥ 20 U/mL.
Time Frame: 4 weeks after the third dose
Population: Evaluated in a subset who got 3 primary doses, had postdose immunogenicity data with no major protocol deviations.For each Ag in the pentavalent, RV, OPV vaccines, non-inferiority shown if 2-sided 95% CI for difference in response proportions (PNEUMOSIL-Synflorix) had lower limit >-0.10. For this, pooled PNUEMOSIL data was used as specified in SAP.
Measure: Count of Participants; unit: Participants
Groups:
- Pneumosil: EPI vaccine immune responses after three doses of Pneumosil
- Synflorix: EPI vaccine immune responses after three doses of Synflorix
Arm/Group | Pneumosil | Synflorix
Number analyzed (Participants) | 447 | 225
Participants
  Anti-Diphtheria Toxoid ≥ 0.1 IU/mL | 447 | 225
  Anti-Tetanus Toxoid ≥ 0.1 IU/mL | 447 | 225
  Anti-HBsAg concentration ≥ 10 mIU/mL | 447 | 224
  Anti-PRP concentration ≥ 0.15 μg/mL | 441 | 224
  Anti-Polio titer ≥ 1:8 (type 1) | 446 | 225
  Anti-Polio titer ≥ 1:8 (type 2) | 374 | 182
  Anti-Polio titer ≥ 1:8 (type 3) | 437 | 222
  Anti-Rotavirus concentration ≥ 20 U/mL | 122 | 61
Statistical Analysis 1: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — Non-inferiority was to be shown if the lower limit of the 95% CI exceeded -10% (for comparisons based on the difference in proportions of antibody responders to EPI vaccines between PNEUMOSIL and Synflorix); Absolute difference for diphtheria = 0.0 — CI could not be computed due to 100% response rate
Statistical Analysis 2: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Absolute difference for Tetanus = 0.0 — CI could not be computed due to 100% response rate
Statistical Analysis 3: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Absolute difference for Hepatitis B = 0.4, 95% CI 2-sided [-0.4 to 2.5]
Statistical Analysis 4: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Absolute difference for Hib = -0.9, 95% CI 2-sided [-2.5 to 1.2]
Statistical Analysis 5: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Absolute difference for Polio type 1 = -0.2, 95% CI 2-sided [-1.3 to 1.5]
Statistical Analysis 6: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Absolute difference for Polio type 2 = 2.8, 95% CI 2-sided [-3.2 to 9.3]
Statistical Analysis 7: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Absolute difference for Polio type 3 = -0.9, 95% CI 2-sided [-3.0 to 1.8]
Statistical Analysis 8: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Absolute difference for Rotavirus = 0.2, 95% CI 2-sided [-7.1 to 7.1]

5. Primary Outcome: Anti-pertussis Toxoid GMCs for the Pertussis Antigen
Description: Anti-pertussis toxoid GMCs for the pertussis antigen
Time Frame: 4 weeks after the third dose
Population: Evaluated in a subset who got 3 primary doses, had postdose immunogenicity data with no major protocol deviations.Non-inferiority was defined as 2-sided 95% CI for the GMC ratio (PNEUMOSIL/Synflorix) with lower limit>0.5 for each of 2 separate antigens (pertussis toxoid and fimbriae).For this analysis, pooled PNUEMOSIL data used as specified in SAP
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Pneumosil | Synflorix
Number analyzed (Participants) | 447 | 225
IU/mL | 50.95 [43.13 to 60.20] | 61.82 [49.58 to 77.09]
Statistical Analysis 1: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — Non-inferiority was to be shown if the lower limit of the 95% CI for the GMC ratio exceeded 0.5 (for pertussis antigens); GMC Ratio for anti-pertussis toxoid = 0.82, 95% CI 2-sided [0.62 to 1.09]

6. Primary Outcome: Anti Fimbriae 2/3 IgG GMCs for the Pertussis Antigen
Description: Anti fimbriae 2/3 IgG GMCs for the pertussis antigen
Time Frame: 4 weeks after the third dose
Population: Evaluated in a subset of subjects who received all primary series doses, had postdose immunogenicity results with no major protocol deviations. Non-inferiority was defined as a two-sided 95% CI for the GMC ratio (PNEUMOSIL/Synflorix) with lower limit > 0.5 for each of 2 separate antigens (pertussis toxoid and fimbriae).
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Pneumosil | Synflorix
Number analyzed (Participants) | 447 | 225
U/mL | 317.97 [275.91 to 366.45] | 324.87 [267.34 to 394.78]
Statistical Analysis 1: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; GMC Ratio for anti-fimbriae 2/3 = 0.98, 95% CI 2-sided [0.77 to 1.25]

7. Primary Outcome: Number and Percentage of Solicited Local and Systemic Reactogenicity by Severity- Vaccination 1
Description: In the primary reactogenicity cohort, local and systemic reactogenicity of the study vaccine was evaluated through day 6 for severity by toxicity grading scale (0 [none], 1 [mild], 2 [moderate], 3 [severe], 4 [life threatening].
Time Frame: 7 days (including day of vaccination)
Population: Sample size for evaluation of solicited local and systemic AEs was approx. 1,125. Evaluated in a subset of subjects who got a study vaccine and had some post-vaccination safety data. Lotwise data was used for clinical lot equivalence evaluation, for safety analyses pooled PNUEMOSIL data was used as specified in SAP.
Measure: Count of Participants; unit: Participants
Groups:
- Pneumosil: Subjects who have received one dose of Pneumosil vaccine
- Synflorix: Subjects who have received one dose of Synflorix vaccine
Arm/Group | Pneumosil | Synflorix
Number analyzed (Participants) | 751 | 364
Participants
  Temperature: Grade 0 | 516 | 249
  Temperature: Grade 1 | 183 | 88
  Temperature: Grade 2 | 52 | 27
  Cutaneous Rash: Grade 0 | 731 | 353
  Cutaneous Rash: Grade 1 | 19 | 10
  Cutaneous Rash: Grade 2 | 1 | 1
  Irritability: Grade 0 | 619 | 301
  Irritability: Grade 1 | 127 | 57
  Irritability: Grade 2 | 5 | 6
  Drowsiness: Grade 0 | 732 | 352
  Drowsiness: Grade 1 | 19 | 12
  Drowsiness: Grade 2 | 0 | 0
  Decreased Appetite: Grade 0 | 728 | 349
  Decreased Appetite: Grade 1 | 22 | 12
  Decreased Appetite: Grade 2 | 1 | 3
  Tenderness: Grade 0 | 539 | 251
  Tenderness: Grade 1 | 185 | 93
  Tenderness: Grade 2 | 27 | 20
  Erythema/Redness: Grade 0 | 736 | 350
  Erythema/Redness: Grade 1 | 15 | 13
  Erythema/Redness: Grade 2 | 0 | 1
  Induration/Swelling: Grade 0 | 731 | 345
  Induration/Swelling: Grade 1 | 17 | 16
  Induration/Swelling: Grade 2 | 3 | 3

8. Primary Outcome: Number and Percentage of Solicited Local and Systemic Reactogenicity by Severity- Vaccination 2
Description: as for outcome 7
Time Frame: 7 days (including day of vaccination)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Groups:
- Pneumosil: Subjects who have received two doses of Pneumosil vaccine
- Synflorix: Subjects who have received two doses of Synflorix vaccine
Arm/Group | Pneumosil | Synflorix
Number analyzed (Participants) | 739 | 361
Participants
  Temperature: Grade 0 | 590 | 271
  Temperature: Grade 1 | 121 | 70
  Temperature: Grade 2 | 25 | 19
  Temperature: Grade 3 | 3 | 1
  Cutaneous Rash: Grade 0 | 727 | 355
  Cutaneous Rash: Grade 1 | 10 | 4
  Cutaneous Rash: Grade 2 | 2 | 1
  Cutaneous Rash: Grade 3 | 0 | 1
  Irritability: Grade 0 | 646 | 324
  Irritability: Grade 1 | 84 | 36
  Irritability: Grade 2 | 8 | 1
  Irritability: Grade 3 | 1 | 0
  Drowsiness: Grade 0 | 726 | 359
  Drowsiness: Grade 1 | 13 | 2
  Drowsiness: Grade 2 | 0 | 0
  Drowsiness: Grade 3 | 0 | 0
  Decreased Appetite: Grade 0 | 728 | 354
  Decreased Appetite: Grade 1 | 10 | 4
  Decreased Appetite: Grade 2 | 0 | 3
  Decreased Appetite: Grade 3 | 1 | 0
  Tenderness: Grade 0 | 585 | 283
  Tenderness: Grade 1 | 127 | 63
  Tenderness: Grade 2 | 27 | 15
  Tenderness: Grade 3 | 0 | 0
  Erythema/Redness: Grade 0 | 725 | 356
  Erythema/Redness: Grade 1 | 14 | 5
  Erythema/Redness: Grade 2 | 0 | 0
  Erythema/Redness: Grade 3 | 0 | 0
  Induration/Swelling: Grade 0 | 724 | 348
  Induration/Swelling: Grade 1 | 14 | 11
  Induration/Swelling: Grade 2 | 1 | 2
  Induration/Swelling: Grade 3 | 0 | 0

9. Primary Outcome: Number and Percentage of Solicited Local and Systemic Reactogenicity by Severity- Vaccination 3
Description: as for outcome 7
Time Frame: 7 days (including day of vaccination)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Groups:
- Pneumosil: Subjects who have received three doses of Pneumosil vaccine
- Synflorix: Subjects who have received three doses of Synflorix vaccine
Arm/Group | Pneumosil | Synflorix
Number analyzed (Participants) | 735 | 360
Participants
  Temperature: Grade 0 | 576 | 301
  Temperature: Grade 1 | 122 | 51
  Temperature: Grade 2 | 37 | 7
  Temperature: Grade 3 | 0 | 1
  Temperature: Grade 4 | 0 | 0
  Cutaneous Rash: Grade 0 | 726 | 358
  Cutaneous Rash: Grade 1 | 9 | 2
  Cutaneous Rash: Grade 2 | 0 | 0
  Cutaneous Rash: Grade 3 | 0 | 0
  Cutaneous Rash: Grade 4 | 0 | 0
  Irritability: Grade 0 | 657 | 316
  Irritability: Grade 1 | 74 | 41
  Irritability: Grade 2 | 3 | 3
  Irritability: Grade 3 | 0 | 0
  Irritability: Grade 4 | 1 | 0
  Drowsiness: Grade 0 | 717 | 352
  Drowsiness: Grade 1 | 17 | 8
  Drowsiness: Grade 2 | 0 | 0
  Drowsiness: Grade 3 | 1 | 0
  Drowsiness: Grade 4 | 0 | 0
  Decreased Appetite: Grade 0 | 716 | 353
  Decreased Appetite: Grade 1 | 17 | 6
  Decreased Appetite: Grade 2 | 1 | 0
  Decreased Appetite: Grade 3 | 1 | 1
  Decreased Appetite: Grade 4 | 0 | 0
  Tenderness: Grade 0 | 605 | 296
  Tenderness: Grade 1 | 110 | 55
  Tenderness: Grade 2 | 20 | 9
  Tenderness: Grade 3 | 0 | 0
  Tenderness: Grade 4 | 0 | 0
  Erythema/Redness: Grade 0 | 730 | 357
  Erythema/Redness: Grade 1 | 4 | 3
  Erythema/Redness: Grade 2 | 1 | 0
  Erythema/Redness: Grade 3 | 0 | 0
  Erythema/Redness: Grade 4 | 0 | 0
  Induration/Swelling: Grade 0 | 727 | 353
  Induration/Swelling: Grade 1 | 7 | 6
  Induration/Swelling: Grade 2 | 1 | 1
  Induration/Swelling: Grade 3 | 0 | 0
  Induration/Swelling: Grade 4 | 0 | 0

10. Primary Outcome: Number and Percentage of Solicited Local and Systemic Reactogenicity by Severity- Booster
Description: as for outcome 7
Time Frame: 7 days (including day of vaccination)
Population: Reported in a subset of subjects who got 3 doses and booster dose of the study vaccine and had post-vaccination safety data.Treatment groups (PNUEMOSIL or Synflorix) were based on actual treatment received at Visit 1. Lotwise data was used for clinical lot equivalence evaluation, for safety analyses pooled PNUEMOSIL data was used (specified in SAP)
Measure: Count of Participants; unit: Participants
Groups:
- Pneumosil: Three doses + 1 booster dose of Pneumosil
- Synflorix: Three doses + 1 booster dose of Synflorix
Arm/Group | Pneumosil | Synflorix
Number analyzed (Participants) | 428 | 213
Participants
  Temperature: Grade 0 | 404 | 197
  Temperature: Grade 1 | 14 | 12
  Temperature: Grade 2 | 9 | 4
  Temperature: Grade 3 | 1 | 0
  Cutaneous Rash: Grade 0 | 424 | 211
  Cutaneous Rash: Grade 1 | 4 | 2
  Cutaneous Rash: Grade 2 | 0 | 0
  Cutaneous Rash: Grade 3 | 0 | 0
  Irritability: Grade 0 | 415 | 207
  Irritability: Grade 1 | 12 | 6
  Irritability: Grade 2 | 1 | 0
  Irritability: Grade 3 | 0 | 0
  Drowsiness: Grade 0 | 418 | 208
  Drowsiness: Grade 1 | 9 | 5
  Drowsiness: Grade 2 | 0 | 0
  Drowsiness: Grade 3 | 1 | 0
  Decreased Appetite: Grade 0 | 425 | 211
  Decreased Appetite: Grade 1 | 2 | 2
  Decreased Appetite: Grade 2 | 1 | 0
  Decreased Appetite: Grade 3 | 0 | 0
  Tenderness: Grade 0 | 395 | 200
  Tenderness: Grade 1 | 28 | 9
  Tenderness: Grade 2 | 5 | 4
  Tenderness: Grade 3 | 0 | 0
  Erythema/Redness: Grade 0 | 428 | 213
  Erythema/Redness: Grade 1 | 0 | 0
  Erythema/Redness: Grade 2 | 0 | 0
  Erythema/Redness: Grade 3 | 0 | 0
  Induration/Swelling: Grade 0 | 423 | 209
  Induration/Swelling: Grade 1 | 5 | 4
  Induration/Swelling: Grade 2 | 0 | 0
  Induration/Swelling: Grade 3 | 0 | 0

11. Primary Outcome: Number and Percentage of All AEs Including SAEs Occurring in Greater Than 1% Subjects by Severity and Relatedness
Description: All subjects were followed up for AEs till 4 weeks post vaccination dose 3 and subjects in the booster cohort were followed up for AEs till 4 weeks post booster vaccination
Time Frame: 4 weeks post last vaccination
Population: Evaluated in all subjects who received a study vaccination and provided some post-vaccination safety data. Treatment groups (PNUEMOSIL or Synflorix) were based on actual treatment received at Visit 1. Lotwise data was used for clinical lot equivalence evaluation, for safety analyses pooled PNUEMOSIL data was used as specified in SAP.
Measure: Count of Participants; unit: Participants
Groups:
- Pneumosil: Primary series who have received three doses and booster cohort who have received three doses + a booster dose of Pneumosil
- Synflorix: Primary series who have received three doses and booster cohort who have received three doses + a booster dose of Synflorix
Arm/Group | Pneumosil | Synflorix
Number analyzed (Participants) | 1503 | 747
Participants
  Upper respiratory tract infection: Mild-Related | 0 | 0
  Upper respiratory tract infection: Mild-Not related | 714 | 366
  Upper respiratory tract infection: Moderate-Related | 0 | 0
  Upper respiratory tract infection: Moderate-Not related | 48 | 26
  Upper respiratory tract infection: Severe-Related | 0 | 0
  Upper respiratory tract infection: Severe-Not related | 2 | 0
  Upper respiratory tract infection: None | 739 | 355
  Furuncle: Mild-Related | 0 | 0
  Furuncle: Mild-Not related | 142 | 62
  Furuncle: Moderate-Related | 0 | 0
  Furuncle: Moderate-Not related | 11 | 3
  Furuncle: Severe-Related | 0 | 0
  Furuncle: Severe-Not related | 0 | 0
  Furuncle: None | 1350 | 682
  Gastroenteritis: Mild-Related | 0 | 0
  Gastroenteritis: Mild-Not related | 125 | 67
  Gastroenteritis: Moderate-Related | 0 | 0
  Gastroenteritis: Moderate-Not related | 27 | 7
  Gastroenteritis: Severe-Related | 0 | 0
  Gastroenteritis: Severe-Not related | 5 | 3
  Gastroenteritis: None | 1346 | 670
  Conjunctivitis: Mild-Related | 0 | 0
  Conjunctivitis: Mild-Not related | 103 | 62
  Conjunctivitis: Moderate-Related | 0 | 0
  Conjunctivitis: Moderate-Not related | 8 | 2
  Conjunctivitis: Severe-Related | 0 | 0
  Conjunctivitis: Severe-Not related | 0 | 0
  Conjunctivitis: None | 1392 | 683
  Bronchiolitis: Mild-Related | 0 | 0
  Bronchiolitis: Mild-Not related | 30 | 32
  Bronchiolitis: Moderate-Related | 0 | 0
  Bronchiolitis: Moderate-Not related | 20 | 8
  Bronchiolitis: Severe-Related | 0 | 0
  Bronchiolitis: Severe-Not related | 13 | 4
  Bronchiolitis: None | 1440 | 703
  Tinea infection: Mild-Related | 0 | 0
  Tinea infection: Mild-Not related | 59 | 21
  Tinea infection: Moderate-Related | 0 | 0
  Tinea infection: Moderate-Not related | 3 | 1
  Tinea infection: Severe-Related | 0 | 0
  Tinea infection: Severe-Not related | 0 | 0
  Tinea infection: None | 1441 | 725
  Febrile infection: Mild-Related | 0 | 0
  Febrile infection: Mild-Not related | 44 | 20
  Febrile infection: Moderate-Related | 0 | 0
  Febrile infection: Moderate-Not related | 9 | 7
  Febrile infection: Severe-Related | 0 | 0
  Febrile infection: Severe-Not related | 0 | 1
  Febrile infection: None | 1450 | 719
  Pneumonia: Mild-Related | 0 | 0
  Pneumonia: Mild-Not related | 17 | 10
  Pneumonia: Moderate-Related | 0 | 0
  Pneumonia: Moderate-Not related | 21 | 5
  Pneumonia: Severe-Related | 0 | 0
  Pneumonia: Severe-Not related | 5 | 6
  Pneumonia: None | 1460 | 726
  Tinea capitis: Mild-Related | 0 | 0
  Tinea capitis: Mild-Not related | 29 | 22
  Tinea capitis: Moderate-Related | 0 | 0
  Tinea capitis: Moderate-Not related | 0 | 0
  Tinea capitis: Severe-Related | 0 | 0
  Tinea capitis: Severe-Not related | 0 | 0
  Tinea capitis: None | 1474 | 725
  Oral candidiasis: Mild-Related | 0 | 0
  Oral candidiasis: Mild-Not related | 31 | 15
  Oral candidiasis: Moderate-Related | 0 | 0
  Oral candidiasis: Moderate-Not related | 4 | 0
  Oral candidiasis: Severe-Related | 0 | 0
  Oral candidiasis: Severe-Not related | 0 | 0
  Oral candidiasis: None | 1468 | 732
  Body tinea: Mild-Related | 0 | 0
  Body tinea: Mild-Not related | 27 | 18
  Body tinea: Moderate-Related | 0 | 0
  Body tinea: Moderate-Not related | 2 | 0
  Body tinea: Severe-Related | 0 | 0
  Body tinea: Severe-Not related | 0 | 0
  Body tinea: None | 1474 | 729
  Impetigo: Mild-Related | 0 | 0
  Impetigo: Mild-Not related | 24 | 19
  Impetigo: Moderate-Related | 0 | 0
  Impetigo: Moderate-Not related | 3 | 0
  Impetigo: Severe-Related | 0 | 0
  Impetigo: Severe-Not related | 0 | 0
  Impetigo: None | 1476 | 728
  Rash pustular: Mild-Related | 0 | 0
  Rash pustular: Mild-Not related | 25 | 15
  Rash pustular: Moderate-Related | 0 | 0
  Rash pustular: Moderate-Not related | 0 | 1
  Rash pustular: Severe-Related | 0 | 0
  Rash pustular: Severe-Not related | 0 | 0
  Rash pustular: None | 1478 | 731
  Skin candida: Mild-Related | 0 | 0
  Skin candida: Mild-Not related | 14 | 11
  Skin candida: Moderate-Related | 0 | 0
  Skin candida: Moderate-Not related | 0 | 0
  Skin candida: Severe-Related | 0 | 0
  Skin candida: Severe-Not related | 0 | 0
  Skin candida: None | 1489 | 736
  Diarrhoea: Mild-Related | 1 | 0
  Diarrhoea: Mild-Not related | 268 | 130
  Diarrhoea: Moderate-Related | 0 | 0
  Diarrhoea: Moderate-Not related | 16 | 3
  Diarrhoea: Severe-Related | 0 | 0
  Diarrhoea: Severe-Not related | 0 | 0
  Diarrhoea: None | 1218 | 614
  Vomiting: Mild-Related | 0 | 1
  Vomiting: Mild-Not related | 22 | 12
  Vomiting: Moderate-Related | 0 | 0
  Vomiting: Moderate-Not related | 2 | 0
  Vomiting: Severe-Related | 0 | 0
  Vomiting: Severe-Not related | 1 | 0
  Vomiting: None | 1478 | 734
  Dermatitis diaper: Mild-Related | 0 | 0
  Dermatitis diaper: Mild-Not related | 34 | 27
  Dermatitis diaper: Moderate-Related | 0 | 0
  Dermatitis diaper: Moderate-Not related | 2 | 1
  Dermatitis diaper: Severe-Related | 0 | 0
  Dermatitis diaper: Severe-Not related | 0 | 0
  Dermatitis diaper: None | 1467 | 719
  Rash maculo-papular: Mild-Related | 0 | 1
  Rash maculo-papular: Mild-Not related | 37 | 14
  Rash maculo-papular: Moderate-Related | 0 | 0
  Rash maculo-papular: Moderate-Not related | 0 | 2
  Rash maculo-papular: Severe-Related | 0 | 0
  Rash maculo-papular: Severe-Not related | 0 | 0
  Rash maculo-papular: None | 1466 | 730
  Rash papular: Mild-Related | 1 | 0
  Rash papular: Mild-Not related | 19 | 11
  Rash papular: Moderate-Related | 0 | 0
  Rash papular: Moderate-Not related | 0 | 0
  Rash papular: Severe-Related | 0 | 0
  Rash papular: Severe-Not related | 0 | 0
  Rash papular: None | 1483 | 736
  Dermatitis contact: Mild-Related | 0 | 0
  Dermatitis contact: Mild-Not related | 16 | 7
  Dermatitis contact: Moderate-Related | 0 | 0
  Dermatitis contact: Moderate-Not related | 2 | 0
  Dermatitis contact: Severe-Related | 0 | 0
  Dermatitis contact: Severe-Not related | 0 | 0
  Dermatitis contact: None | 1485 | 740
  Dermatitis atopic: Mild-Related | 0 | 0
  Dermatitis atopic: Mild-Not related | 12 | 10
  Dermatitis atopic: Moderate-Related | 0 | 0
  Dermatitis atopic: Moderate-Not related | 0 | 1
  Dermatitis atopic: Severe-Related | 0 | 0
  Dermatitis atopic: Severe-Not related | 0 | 0
  Dermatitis atopic: None | 1491 | 736
  Seborrhoeic dermatitis: Mild-Related | 0 | 0
  Seborrhoeic dermatitis: Mild-Not related | 16 | 5
  Seborrhoeic dermatitis: Moderate-Related | 0 | 0
  Seborrhoeic dermatitis: Moderate-Not related | 1 | 0
  Seborrhoeic dermatitis: Severe-Related | 0 | 0
  Seborrhoeic dermatitis: Severe-Not related | 0 | 0
  Seborrhoeic dermatitis: None | 1486 | 742
  Cough: Mild-Related | 0 | 0
  Cough: Mild-Not related | 95 | 38
  Cough: Moderate-Related | 0 | 0
  Cough: Moderate-Not related | 0 | 1
  Cough: Severe-Related | 0 | 0
  Cough: Severe-Not related | 0 | 0
  Cough: None | 1408 | 708
  Pyrexia: Mild-Related | 1 | 0
  Pyrexia: Mild-Not related | 17 | 15
  Pyrexia: Moderate-Related | 1 | 0
  Pyrexia: Moderate-Not related | 8 | 1
  Pyrexia: Severe-Related | 3 | 0
  Pyrexia: Severe-Not related | 1 | 0
  Pyrexia: None | 1472 | 731
  Thermal burn: Mild-Related | 0 | 0
  Thermal burn: Mild-Not related | 7 | 10
  Thermal burn: Moderate-Related | 0 | 0
  Thermal burn: Moderate-Not related | 2 | 1
  Thermal burn: Severe-Related | 0 | 0
  Thermal burn: Severe-Not related | 0 | 0
  Thermal burn: None | 1494 | 736

12. Primary Outcome: Number and Percentage of All SAEs by Severity and Relatedness
Description: All subjects were followed up for SAEs till 4 weeks post vaccination dose 3 and subjects in the booster cohort were followed up for SAEs till 4 weeks post booster vaccination
Time Frame: 4 weeks post last vaccination
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Pneumosil | Synflorix
Number analyzed (Participants) | 1503 | 747
Participants
  Bronchiolitis: Moderate-Not Related | 0 | 0
  Bronchiolitis: Severe-Not Related | 13 | 4
  Bronchiolitis: None | 1490 | 743
  Gastroenteritis: Moderate-Not Related | 4 | 0
  Gastroenteritis: Severe-Not Related | 5 | 3
  Gastroenteritis: None | 1494 | 744
  Pneumonia: Moderate-Not Related | 0 | 0
  Pneumonia: Severe-Not Related | 4 | 6
  Pneumonia: None | 1499 | 741
  Dysentery: Moderate-Not Related | 0 | 0
  Dysentery: Severe-Not Related | 0 | 1
  Dysentery: None | 1503 | 746
  Febrile infection: Moderate-Not Related | 0 | 1
  Febrile infection: Severe-Not Related | 0 | 0
  Febrile infection: None | 1503 | 746
  HIV infection WHO clinical stage IV: Moderate-Not Related | 0 | 0
  HIV infection WHO clinical stage IV: Severe-Not Related | 0 | 1
  HIV infection WHO clinical stage IV: None | 1503 | 746
  Meningitis pneumococcal: Moderate-Not Related | 0 | 0
  Meningitis pneumococcal: Severe-Not Related | 1 | 0
  Meningitis pneumococcal: None | 1502 | 747
  Perinatal HIV infection: Moderate-Not Related | 0 | 0
  Perinatal HIV infection: Severe-Not Related | 0 | 1
  Perinatal HIV infection: None | 1503 | 746
  Periorbital cellulitis: Moderate-Not Related | 0 | 0
  Periorbital cellulitis: Severe-Not Related | 0 | 1
  Periorbital cellulitis: None | 1503 | 746
  Upper respiratory tract infection: Moderate-Not Related | 0 | 0
  Upper respiratory tract infection: Severe-Not Related | 1 | 0
  Upper respiratory tract infection: None | 1502 | 747
  Fallot's tetralogy: Moderate-Not Related | 0 | 0
  Fallot's tetralogy: Severe-Not Related | 1 | 1
  Fallot's tetralogy: None | 1502 | 746
  Trisomy 21: Moderate-Not Related | 0 | 0
  Trisomy 21: Severe-Not Related | 2 | 0
  Trisomy 21: None | 1501 | 747
  Atrioventricular septal defect: Moderate-Not Related | 0 | 0
  Atrioventricular septal defect: Severe-Not Related | 1 | 0
  Atrioventricular septal defect: None | 1502 | 747
  Intussusception: Moderate-Not Related | 0 | 0
  Intussusception: Severe-Not Related | 2 | 0
  Intussusception: None | 1501 | 747
  Diarrhoea haemorrhagic: Moderate-Not Related | 0 | 0
  Diarrhoea haemorrhagic: Severe-Not Related | 1 | 0
  Diarrhoea haemorrhagic: None | 1502 | 747
  Vomiting: Moderate-Not Related | 0 | 0
  Vomiting: Severe-Not Related | 1 | 0
  Vomiting: None | 1502 | 747
  Developmental delay: Moderate-Not Related | 0 | 0
  Developmental delay: Severe-Not Related | 1 | 0
  Developmental delay: None | 1502 | 747
  Malnutrition: Moderate-Not Related | 0 | 0
  Malnutrition: Severe-Not Related | 0 | 1
  Malnutrition: None | 1503 | 746
  Seizure: Moderate-Not Related | 0 | 0
  Seizure: Severe-Not Related | 1 | 0
  Seizure: None | 1502 | 747
  Epistaxis: Moderate-Not Related | 0 | 0
  Epistaxis: Severe-Not Related | 1 | 0
  Epistaxis: None | 1502 | 747
  Stevens-Johnson syndrome: Moderate-Not Related | 0 | 0
  Stevens-Johnson syndrome: Severe-Not Related | 1 | 0
  Stevens-Johnson syndrome: None | 1502 | 747

13. Secondary Outcome: Number and Percentage of Subjects With 6A and 19A Serotype-specific Concentrations of Immunoglobulin G Antibody
Description: Subjects with 6A and 19A serotype-specific concentrations of immunoglobulin G (IgG) antibody measured by ELISA
Time Frame: 4 weeks after the third dose
Population: For 6A and 19A serotypes, proportions with IgG concentration ≥ 0.35 µg/mL were compared using a z-test for proportions.Test was done at the 2-sided 2.5% significance level to adjust for superiority test. Analysis was done on pooled PNEUMOSIL data as specified in SAP
Measure: Count of Participants; unit: Participants
Arm/Group | Pneumosil | Synflorix
Number analyzed (Participants) | 1458 | 724
Participants
  Pn IgG Type 6A | 1193 | 62
  Pn IgG Type 19A: number analyzed (Participants) | 1454 | 721
  Pn IgG Type 19A | 1386 | 293
Statistical Analysis 1: Comparison: Pneumosil vs Synflorix; Test type: Superiority — Proportions with IgG concentration ≥ 0.35 µg/mL will be compared using a z-test for proportions. The test will be done at the two-sided 2.5% significance level to adjust for the two superiority tests. 97.5% CIs for treatment-group differences in response, will also be reported; Difference for Type 6A = 73.3, 97.5% CI 2-sided [69.8 to 76.3]
Statistical Analysis 2: Comparison: Pneumosil vs Synflorix; Test type: Superiority — [test comment as in outcome 13, analysis 1]; Difference for Type 19A = 54.7, 97.5% CI 2-sided [50.3 to 58.9]

14. Secondary Outcome: 6A and 19A Serotype Specific Geometric Mean Concentration of IgG Antibody
Description: 6A and 19A Serotype Specific Immune Responses in terms of IgG GMCs measured by ELISA
Time Frame: 4 weeks after the third dose
Population: For 6A and 19A serotypes, GMCs were compared by a two-sample t-test on the difference.Test was done at the 2-sided 2.5% significance level to adjust for superiority test.The 95% CIs around treatment-group responses, and 97.5% CIs for treatment-group differences in response were reported.Analysis was done on pooled PNEUMOSIL data as specified in SAP
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Pneumosil | Synflorix
Number analyzed (Participants) | 1458 | 724
µg/mL
  Pn IgG Type 6A | 1.00 [0.95 to 1.06] | 0.12 [0.11 to 0.12]
  Pn IgG Type 19A: number analyzed (Participants) | 1454 | 721
  Pn IgG Type 19A | 1.64 [1.57 to 1.72] | 0.29 [0.27 to 0.31]
Statistical Analysis 1: Comparison: Pneumosil vs Synflorix; Test type: Superiority — For each of the two serotypes, GMCs are compared by a two-sample t-test on the difference between means of log10 (antibody). The test was done at the two-sided 2.5% significance level to adjust for the two superiority tests. 97.5% CIs for treatment-group differences in response, are also be reported; Pn IgG type 6A GMC Ratio = 8.51, 97.5% CI 2-sided [7.68 to 9.43]
Statistical Analysis 2: Comparison: Pneumosil vs Synflorix; Test type: Superiority — [test comment as in outcome 14, analysis 1]; Pn IgG type 19A GMC Ratio = 5.64, 97.5% CI 2-sided [5.14 to 6.18]

15. Secondary Outcome: Number and Percentage of Subjects With Functional Antibody Responses
Description: Serotype-specific functional antibody titer measured by OPA
Time Frame: 4 weeks after the third dose
Population: In a subset of subjects who got 3 primary doses of study vaccines, had postdose immunogenicity measurement and no major protocol deviations, functional immune responses induced by PNEUMOSIL were compared to Synflorix for 10 serotypes in PNEUMOSIL, i.e., OPA seroresponse rate (titer≥1:8) differences.Pooled PNEUMOSIL data was used as noted in the SAP
Measure: Count of Participants; unit: Participants
Arm/Group | Pneumosil | Synflorix
Number analyzed (Participants) | 247 | 250
Participants
  OPA Type 1: number analyzed (Participants) | 247 | 249
  OPA Type 1 | 229 | 188
  OPA Type 5: number analyzed (Participants) | 247 | 249
  OPA Type 5 | 244 | 239
  OPA Type 6A: number analyzed (Participants) | 247 | 241
  OPA Type 6A | 240 | 36
  OPA Type 6B: number analyzed (Participants) | 243 | 245
  OPA Type 6B | 233 | 212
  OPA Type 7F | 247 | 249
  OPA Type 9V: number analyzed (Participants) | 242 | 249
  OPA Type 9V | 242 | 249
  OPA Type 14: number analyzed (Participants) | 244 | 247
  OPA Type 14 | 237 | 242
  OPA Type 19A: number analyzed (Participants) | 247 | 236
  OPA Type 19A | 228 | 92
  OPA Type 19F | 239 | 246
  OPA Type 23F: number analyzed (Participants) | 246 | 243
  OPA Type 23F | 246 | 243
Statistical Analysis 1: Comparison: Pneumosil vs Synflorix; Test type: Other — Serotype specific functional antibody responses measured by OPA titer to Pneumosil in comparison with Synflorix for each of the 10 serotypes; OPA Type 1 = 17.2, 95% CI 2-sided [11.0 to 23.6]
Statistical Analysis 2: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 15, analysis 1]; OPA Type 5 = 2.8, 95% CI 2-sided [-0.0 to 6.2]
Statistical Analysis 3: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 15, analysis 1]; OPA Type 6A = 82.2, 95% CI 2-sided [76.7 to 86.6]
Statistical Analysis 4: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 15, analysis 1]; OPA Type 6B = 9.4, 95% CI 2-sided [4.5 to 14.6]
Statistical Analysis 5: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 15, analysis 1]; OPA Type 7F = 0.4, 95% CI 2-sided [-1.1 to 2.2]
Statistical Analysis 6: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 15, analysis 1]; OPA Type 9V = 0.0 — CI could not be computed due to 100% response rate
Statistical Analysis 7: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 15, analysis 1]; OPA Type14 = -0.8, 95% CI 2-sided [-4.0 to 2.2]
Statistical Analysis 8: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 15, analysis 1]; OPA Type 19A = 53.3, 95% CI 2-sided [46.0 to 60.1]
Statistical Analysis 9: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 15, analysis 1]; OPA Type 19F = -1.6, 95% CI 2-sided [-4.9 to 1.2]
Statistical Analysis 10: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 15, analysis 1]; OPA Type 23F = 0.0 — CI could not be computed due to 100% response rate

16. Secondary Outcome: Serotype-specific OPA Geometric Mean Titer
Description: Serotype-specific functional antibody titer measured by OPA and expressed as OPA GMT in a subset
Time Frame: 4 weeks after the third dose
Population: In a subset of subjects who got 3 primary doses of study vaccines, had postdose immunogenicity measurement and no major protocol deviations, functional immune responses induced by PNEUMOSIL were compared to Synflorix for 10 serotypes in PNEUMOSIL, i.e., ratio of OPA GMTs (and corresponding 95% CIs).Pooled PNEUMOSIL data was used as noted in the SAP
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Pneumosil | Synflorix
Number analyzed (Participants) | 247 | 250
titer
  OPA Type 1: number analyzed (Participants) | 247 | 249
  OPA Type 1 | 85.17 [71.34 to 101.69] | 27.55 [22.96 to 33.06]
  OPA Type 5: number analyzed (Participants) | 247 | 249
  OPA Type 5 | 161.34 [139.94 to 186.02] | 115.93 [98.85 to 135.97]
  OPA Type 6A: number analyzed (Participants) | 247 | 241
  OPA Type 6A | 1317.16 [1109.36 to 1563.88] | 7.06 [5.83 to 8.56]
  OPA Type 6B: number analyzed (Participants) | 243 | 245
  OPA Type 6B | 913.52 [745.97 to 1118.70] | 467.65 [365.27 to 598.73]
  OPA Type 7F | 1833.71 [1612.31 to 2085.51] | 1586.75 [1392.62 to 1807.94]
  OPA Type 9V: number analyzed (Participants) | 242 | 249
  OPA Type 9V | 141.72 [113.36 to 177.16] | 376.77 [324.01 to 438.13]
  OPA Type 14: number analyzed (Participants) | 244 | 247
  OPA Type 14 | 1019.34 [816.53 to 1272.52] | 1102.64 [878.56 to 1383.87]
  OPA 19A: number analyzed (Participants) | 247 | 236
  OPA 19A | 148.59 [121.35 to 181.95] | 11.09 [9.19 to 13.39]
  OPA 19F | 594.27 [509.98 to 692.49] | 895.39 [784.96 to 1021.35]
  OPA 23F: number analyzed (Participants) | 246 | 243
  OPA 23F | 767.24 [648.95 to 907.10] | 253.09 [197.10 to 325.00]
Statistical Analysis 1: Comparison: Pneumosil vs Synflorix; Test type: Other — Serotype specific functional antibody responses measured by OPA to Pneumosil in comparison with Synflorix for each of the 10 serotypes (GMT Ratio); OPA GMT Ratio-Type 1 = 3.09, 95% CI 2-sided [2.40 to 3.98]
Statistical Analysis 2: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 16, analysis 1]; OPA GMT Ratio-Type 5 = 1.39, 95% CI 2-sided [1.12 to 1.72]
Statistical Analysis 3: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 16, analysis 1]; OPA GMT Ratio-Type 6A = 186, 95% CI 2-sided [144 to 241]
Statistical Analysis 4: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 16, analysis 1]; OPA GMT Ratio-Type 6B = 1.95, 95% CI 2-sided [1.42 to 2.69]
Statistical Analysis 5: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 16, analysis 1]; OPA GMT Ratio-Type 7F = 1.16, 95% CI 2-sided [0.96 to 1.39]
Statistical Analysis 6: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 16, analysis 1]; OPA GMT Ratio-Type 9V = 0.38, 95% CI 2-sided [0.29 to 0.49]
Statistical Analysis 7: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 16, analysis 1]; OPA GMT Ratio-Type 14 = 0.92, 95% CI 2-sided [0.67 to 1.27]
Statistical Analysis 8: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 16, analysis 1]; OPA GMT Ratio-Type 19A = 13.4, 95% CI 2-sided [10.2 to 17.7]
Statistical Analysis 9: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 16, analysis 1]; OPA GMT Ratio-Type 19F = 0.66, 95% CI 2-sided [0.54 to 0.81]
Statistical Analysis 10: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 16, analysis 1]; OPA GMT Ratio-Type 23F = 3.03, 95% CI 2-sided [2.25 to 4.09]

17. Secondary Outcome: Comparison of Serotype-specific Geometric Mean Concentration of IgG Antibody Response 4 Weeks After a 3-dose Primary Series to 4 Weeks After a Booster Dose
Description: Comparison of Serotype-specific booster responses (antibody concentrations) measured by ELISA from 4 weeks after a 3-dose primary series to 4 weeks after a booster dose
Time Frame: 4 weeks post booster vaccination
Population: In a subset who got 3 primary series+booster dose of study vaccines, had postdose immunogenicity measurement & no major PDs, comparisons based on ratios of IgG GMC post booster to IgG GMC post primary series. Comparison done using ratios of the ratios for the 2 treatment groups (PNEUMOSIL ratio/Synflorix ratio), & corresponding 95% CIs.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Groups:
- 4 Weeks Post Dose 3-Pneumosil: Three doses of Pneumosil in a subset
- 4 Weeks Post Booster-Pneumosil: Three doses + 1 booster dose of Pneumosil in a subset
- 4 Weeks Post Dose 3-Synflorix: Three doses of Synflorix in a subset
- 4 Weeks Post Booster-Synflorix: Three doses + 1 booster dose of Synflorix in a subset
Arm/Group | 4 Weeks Post Dose 3-Pneumosil | 4 Weeks Post Booster-Pneumosil | 4 Weeks Post Dose 3-Synflorix | 4 Weeks Post Booster-Synflorix
Number analyzed (Participants) | 436 | 425 | 216 | 209
µg/mL
  Pn IgG Type 1: number analyzed (Participants) | 424 | 424 | 208 | 208
  Pn IgG Type 1 | 4.05 [3.76 to 4.36] | 5.71 [5.25 to 6.21] | 2.12 [1.88 to 2.38] | 2.47 [2.19 to 2.80]
  Pn IgG Type 5: number analyzed (Participants) | 424 | 424 | 207 | 207
  Pn IgG Type 5 | 1.49 [1.39 to 1.59] | 1.31 [1.21 to 1.41] | 1.26 [1.14 to 1.38] | 0.84 [0.76 to 0.93]
  Pn IgG Type 6A: number analyzed (Participants) | 423 | 423 | 208 | 208
  Pn IgG Type 6A | 1.09 [0.98 to 1.22] | 4.86 [4.40 to 5.38] | 0.12 [0.11 to 0.14] | 0.42 [0.36 to 0.50]
  Pn IgG Type 6B: number analyzed (Participants) | 422 | 422 | 208 | 208
  Pn IgG Type 6B | 1.29 [1.13 to 1.48] | 8.32 [7.70 to 8.99] | 1.15 [0.94 to 1.41] | 4.44 [4.00 to 4.93]
  Pn IgG Type 7F: number analyzed (Participants) | 424 | 424 | 208 | 208
  Pn IgG Type 7F | 3.12 [2.89 to 3.37] | 6.36 [5.87 to 6.89] | 2.49 [2.22 to 2.79] | 4.07 [3.67 to 4.52]
  Pn IgG Type 9V: number analyzed (Participants) | 423 | 423 | 208 | 208
  Pn IgG Type 9V | 1.29 [1.20 to 1.39] | 1.80 [1.67 to 1.94] | 1.43 [1.28 to 1.60] | 2.08 [1.87 to 2.31]
  Pn IgG Type 14: number analyzed (Participants) | 419 | 419 | 203 | 203
  Pn IgG Type 14 | 5.06 [4.57 to 5.62] | 6.84 [6.08 to 7.68] | 3.86 [3.25 to 4.57] | 4.67 [2.92 to 5.55]
  Pn IgG Type 19A: number analyzed (Participants) | 421 | 421 | 204 | 204
  Pn IgG Type 19A | 1.50 [1.37 to 1.64] | 3.97 [3.63 to 4.33] | 0.26 [0.23 to 0.31] | 0.95 [0.79 to 1.15]
  Pn IgG Type 19F: number analyzed (Participants) | 414 | 414 | 203 | 203
  Pn IgG Type 19F | 4.16 [3.85 to 4.48] | 6.18 [5.70 to 6.71] | 6.31 [5.51 to 7.24] | 9.79 [8.77 to 10.92]
  Pn IgG Type 23F: number analyzed (Participants) | 423 | 423 | 208 | 208
  Pn IgG Type 23F | 1.65 [1.50 to 1.80] | 4.11 [3.75 to 4.50] | 0.94 [0.80 to 1.11] | 2.15 [1.90 to 2.44]
Statistical Analysis 1: Comparison: 4 Weeks Post Dose 3-Pneumosil vs 4 Weeks Post Booster-Pneumosil; Test type: Other — The comparisons were based on the ratio of IgG GMC post-booster to the IgG GMC post-primary series in the Booster Cohort restricted to subjects who contributed relevant data at both time points; Pn IgG type 1 GMC Ratio = 1.41, 95% CI 2-sided [1.31 to 1.52]
Statistical Analysis 2: Comparison: 4 Weeks Post Dose 3-Pneumosil vs 4 Weeks Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 17, analysis 1]; Pn IgG type 5 GMC Ratio = 0.88, 95% CI 2-sided [0.81 to 0.95]
Statistical Analysis 3: Comparison: 4 Weeks Post Dose 3-Pneumosil vs 4 Weeks Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 17, analysis 1]; Pn IgG type 6A GMC Ratio = 4.46, 95% CI 2-sided [4.01 to 4.96]
Statistical Analysis 4: Comparison: 4 Weeks Post Dose 3-Pneumosil vs 4 Weeks Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 17, analysis 1]; Pn IgG type 6B GMC Ratio = 6.43, 95% CI 2-sided [5.70 to 7.26]
Statistical Analysis 5: Comparison: 4 Weeks Post Dose 3-Pneumosil vs 4 Weeks Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 17, analysis 1]; Pn IgG type 7F GMC Ratio = 2.04, 95% CI 2-sided [1.89 to 2.19]
Statistical Analysis 6: Comparison: 4 Weeks Post Dose 3-Pneumosil vs 4 Weeks Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 17, analysis 1]; Pn IgG type 9V GMC Ratio = 1.39, 95% CI 2-sided [1.29 to 1.50]
Statistical Analysis 7: Comparison: 4 Weeks Post Dose 3-Pneumosil vs 4 Weeks Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 17, analysis 1]; Pn IgG type 14 GMC Ratio = 1.35, 95% CI 2-sided [1.21 to 1.51]
Statistical Analysis 8: Comparison: 4 Weeks Post Dose 3-Pneumosil vs 4 Weeks Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 17, analysis 1]; Pn IgG type 19A GMC Ratio = 2.64, 95% CI 2-sided [2.40 to 2.91]
Statistical Analysis 9: Comparison: 4 Weeks Post Dose 3-Pneumosil vs 4 Weeks Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 17, analysis 1]; Pn IgG type 19F GMC Ratio = 1.49, 95% CI 2-sided [1.36 to 1.63]
Statistical Analysis 10: Comparison: 4 Weeks Post Dose 3-Pneumosil vs 4 Weeks Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 17, analysis 1]; Pn IgG type 23F GMC Ratio = 2.50, 95% CI 2-sided [2.29 to 2.72]
Statistical Analysis 11: Comparison: 4 Weeks Post Dose 3-Synflorix vs 4 Weeks Post Booster-Synflorix; Test type: Other — [test comment as in outcome 17, analysis 1]; Pn IgG type 1 GMC Ratio = 1.17, 95% CI 2-sided [1.06 to 1.28]
Statistical Analysis 12: Comparison: 4 Weeks Post Dose 3-Synflorix vs 4 Weeks Post Booster-Synflorix; Test type: Other — [test comment as in outcome 17, analysis 1]; Pn IgG type 5 GMC Ratio = 0.67, 95% CI 2-sided [0.61 to 0.74]
Statistical Analysis 13: Comparison: 4 Weeks Post Dose 3-Synflorix vs 4 Weeks Post Booster-Synflorix; Test type: Other — [test comment as in outcome 17, analysis 1]; Pn IgG type 6A GMC Ratio = 3.49, 95% CI 2-sided [2.97 to 4.11]
Statistical Analysis 14: Comparison: 4 Weeks Post Dose 3-Synflorix vs 4 Weeks Post Booster-Synflorix; Test type: Other — [test comment as in outcome 17, analysis 1]; Pn IgG type 6B GMC Ratio = 3.85, 95% CI 2-sided [3.23 to 4.59]
Statistical Analysis 15: Comparison: 4 Weeks Post Dose 3-Synflorix vs 4 Weeks Post Booster-Synflorix; Test type: Other — [test comment as in outcome 17, analysis 1]; Pn IgG type 7F GMC Ratio = 1.63, 95% CI 2-sided [1.47 to 1.82]
Statistical Analysis 16: Comparison: 4 Weeks Post Dose 3-Synflorix vs 4 Weeks Post Booster-Synflorix; Test type: Other — [test comment as in outcome 17, analysis 1]; Pn IgG type 9V GMC Ratio = 1.46, 95% CI 2-sided [1.31 to 1.62]
Statistical Analysis 17: Comparison: 4 Weeks Post Dose 3-Synflorix vs 4 Weeks Post Booster-Synflorix; Test type: Other — [test comment as in outcome 17, analysis 1]; Pn IgG type 14 GMC Ratio = 1.21, 95% CI 2-sided [1.03 to 1.42]
Statistical Analysis 18: Comparison: 4 Weeks Post Dose 3-Synflorix vs 4 Weeks Post Booster-Synflorix; Test type: Other — [test comment as in outcome 17, analysis 1]; Pn IgG type 19A GMC Ratio = 3.60, 95% CI 2-sided [2.99 to 4.33]
Statistical Analysis 19: Comparison: 4 Weeks Post Dose 3-Synflorix vs 4 Weeks Post Booster-Synflorix; Test type: Other — [test comment as in outcome 17, analysis 1]; Pn IgG type 19F GMC Ratio = 1.55, 95% CI 2-sided [1.38 to 1.75]
Statistical Analysis 20: Comparison: 4 Weeks Post Dose 3-Synflorix vs 4 Weeks Post Booster-Synflorix; Test type: Other — [test comment as in outcome 17, analysis 1]; Pn IgG type 23F GMC Ratio = 2.29, 95% CI 2-sided [1.98 to 2.65]

18. Secondary Outcome: Serotype-specific Geometric Mean Concentration of IgG Antibody Response and Treatment-Group GMC Ratios 4 Weeks After a Booster Dose
Description: Comparison of Serotype-specific booster responses (antibody concentrations) to PNEUMOSIL in comparison to Synflorix 4 weeks after a booster dose
Time Frame: 4 weeks post booster vaccination
Population: In a subset of subjects who got 3 primary series and a booster dose of study vaccines, had postdose immunogenicity measurement(s) with no major protocol deviations, serotype-specific GMC of IgG Antibody and treatment group ratios of IgG GMCs (with corresponding 95% CIs) were evaluated. Pooled PNEUMOSIL data was used for this analysis as per SAP
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Pneumosil | Synflorix
Number analyzed (Participants) | 425 | 209
µg/mL
  Pn IgG Type 1 | 5.73 [5.27 to 6.22] | 2.45 [2.16 to 2.78]
  Pn IgG Type 5: number analyzed (Participants) | 425 | 208
  Pn IgG Type 5 | 1.31 [1.21 to 1.41] | 0.83 [0.75 to 0.92]
  Pn IgG Type 6A: number analyzed (Participants) | 424 | 209
  Pn IgG Type 6A | 4.87 [4.41 to 5.39] | 0.42 [0.35 to 0.49]
  Pn IgG Type 6B: number analyzed (Participants) | 423 | 209
  Pn IgG Type 6B | 8.33 [7.71 to 9.00] | 4.42 [3.98 to 4.90]
  Pn IgG Type 7F | 6.37 [5.88 to 6.90] | 4.06 [3.65 to 4.50]
  Pn IgG Type 9V: number analyzed (Participants) | 424 | 209
  Pn IgG Type 9V | 1.81 [1.67 to 1.95] | 2.07 [1.87 to 2.30]
  Pn IgG Type 14: number analyzed (Participants) | 420 | 204
  Pn IgG Type 14 | 6.85 [6.09 to 7.70] | 4.62 [3.88 to 5.50]
  Pn IgG Type 19A: number analyzed (Participants) | 423 | 205
  Pn IgG Type 19A | 3.97 [3.64 to 4.34] | 0.94 [0.78 to 1.14]
  Pn IgG Type 19F: number analyzed (Participants) | 416 | 204
  Pn IgG Type 19F | 6.16 [5.68 to 6.68] | 9.70 [8.68 to 10.83]
  Pn IgG Type 23F | 4.08 [3.72 to 4.47] | 2.13 [1.88 to 2.42]
Statistical Analysis 1: Comparison: Pneumosil vs Synflorix; Test type: Other — The vaccines were compared using the ratios of the GMC ratios for the two treatment groups, i.e., the PNEUMOSIL ratio divided by the Synflorix ratio, and the corresponding 95% CIs based on log linear random effects models; Pn IgG type 1 GMC Ratio = 2.34, 95% CI 2-sided [2.02 to 2.71]
Statistical Analysis 2: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 18, analysis 1]; Pn IgG type 5 GMC Ratio = 1.57, 95% CI 2-sided [1.38 to 1.79]
Statistical Analysis 3: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 18, analysis 1]; Pn IgG type 6A GMC Ratio = 11.6, 95% CI 2-sided [9.67 to 14.0]
Statistical Analysis 4: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 18, analysis 1]; Pn IgG type 6B GMC Ratio = 1.89, 95% CI 2-sided [1.65 to 2.15]
Statistical Analysis 5: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 18, analysis 1]; Pn IgG type 7F GMC Ratio = 1.57, 95% CI 2-sided [1.37 to 1.80]
Statistical Analysis 6: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 18, analysis 1]; Pn IgG type 9V GMC Ratio = 0.87, 95% CI 2-sided [0.76 to 0.99]
Statistical Analysis 7: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 18, analysis 1]; Pn IgG type 14 GMC Ratio = 1.48, 95% CI 2-sided [1.21 to 1.82]
Statistical Analysis 8: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 18, analysis 1]; Pn IgG type 19A GMC Ratio = 4.22, 95% CI 2-sided [3.52 to 5.06]
Statistical Analysis 9: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 18, analysis 1]; Pn IgG type 19F GMC Ratio = 0.63, 95% CI 2-sided [0.55 to 0.73]
Statistical Analysis 10: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 18, analysis 1]; Pn IgG type 23F GMC Ratio = 1.91, 95% CI 2-sided [1.63 to 2.24]

19. Secondary Outcome: Comparison of Functional Response (OPA) From 4 Weeks After a 3-dose Primary Series to 4 Weeks After a Booster Dose
Description: Comparison of Serotype-specific booster responses (functional response-OPA) from 4 weeks after a 3-dose primary series to 4 weeks after a booster dose
Time Frame: 4 weeks post booster vaccination
Population: In a subset who got 3 primary series+booster dose of study vaccines, had postdose immunogenicity measurement & no major PDs, comparisons based on ratios of OPA GMT post booster to OPA GMT post primary series. Comparison done using ratios of the ratios for the 2 treatment groups (PNEUMOSIL ratio/Synflorix ratio), & corresponding 95% CIs.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 4 Weeks Post Dose 3-Pneumosil | 4 Weeks Post Booster-Pneumosil | 4 Weeks Post Dose 3-Synflorix | 4 Weeks Post Booster-Synflorix
Number analyzed (Participants) | 239 | 99 | 214 | 100
titer
  OPA Type 1: number analyzed (Participants) | 98 | 98 | 97 | 97
  OPA Type 1 | 99.21 [75.22 to 130.9] | 344.5 [261.8 to 453.5] | 29.76 [21.73 to 40.78] | 187.2 [141.6 to 247.4]
  OPA Type 5: number analyzed (Participants) | 99 | 99 | 100 | 100
  OPA Type 5 | 161.2 [126.8 to 205.0] | 409.9 [312.4 to 537.8] | 112.9 [86.79 to 146.9] | 360.6 [281.9 to 461.2]
  OPA Type 6A: number analyzed (Participants) | 98 | 98 | 92 | 92
  OPA Type 6A | 1225 [900.0 to 1666] | 3063 [2329 to 4030] | 6.44 [4.80 to 8.64] | 39.96 [22.94 to 69.59]
  OPA Type 6B: number analyzed (Participants) | 96 | 96 | 98 | 98
  OPA Type 6B | 771.4 [527.2 to 1129] | 2897 [2259 to 3714] | 495.2 [339.6 to 722.1] | 1610 [1271 to 2040]
  OPA Type 7F: number analyzed (Participants) | 99 | 99 | 100 | 100
  OPA Type 7F | 1795 [1461 to 2205] | 6977 [5602 to 8691] | 1438 [1136 to 1820] | 4036 [3270 to 4981]
  OPA Type 9V: number analyzed (Participants) | 95 | 95 | 100 | 100
  OPA Type 9V | 168.7 [117.4 to 242.4] | 1155 [871.4 to 1530] | 417.0 [323.3 to 537.8] | 1229 [979.3 to 1542]
  OPA Type 14: number analyzed (Participants) | 95 | 95 | 98 | 98
  OPA Type 14 | 1254 [885.8 to 1776] | 3069 [2287 to 4118] | 866.8 [579.6 to 1296] | 1401 [967.4 to 2029]
  OPA Type 19A: number analyzed (Participants) | 97 | 97 | 92 | 92
  OPA Type 19A | 177.5 [131.0 to 240.5] | 645.6 [489.7 to 851.0] | 8.89 [6.81 to 11.60] | 53.15 [33.24 to 84.99]
  OPA Type 19F: number analyzed (Participants) | 99 | 99 | 98 | 98
  OPA Type 19F | 669.9 [533.6 to 841.2] | 1592 [1256 to 2019] | 801.0 [624.1 to 1028] | 1580 [1190 to 2099]
  OPA Type 23F: number analyzed (Participants) | 99 | 99 | 94 | 94
  OPA Type 23F | 774.5 [588.3 to 1020] | 3847 [2962 to 4996] | 211.7 [142.0 to 315.7] | 1213 [945.7 to 1557]
Statistical Analysis 1: Comparison: 4 Weeks Post Dose 3-Pneumosil vs 4 Weeks Post Booster-Pneumosil; Test type: Other — The comparisons were based on OPA GMTs 4 weeks post primary series and 4 weeks post booster for the OPA subset of the booster cohort. It was restricted to subjects who contributed relevant data at both time points; OPA GMT Ratio-Type 1 = 3.47, 95% CI 2-sided [2.72 to 4.44]
Statistical Analysis 2: Comparison: 4 Weeks Post Dose 3-Pneumosil vs 4 Weeks Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 19, analysis 1]; OPA GMT Ratio-Type 5 = 2.54, 95% CI 2-sided [2.06 to 3.13]
Statistical Analysis 3: Comparison: 4 Weeks Post Dose 3-Pneumosil vs 4 Weeks Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 19, analysis 1]; OPA GMT Ratio-Type 6A = 2.50, 95% CI 2-sided [1.83 to 3.42]
Statistical Analysis 4: Comparison: 4 Weeks Post Dose 3-Pneumosil vs 4 Weeks Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 19, analysis 1]; OPA GMT Ratio-Type 6B = 3.76, 95% CI 2-sided [2.48 to 5.69]
Statistical Analysis 5: Comparison: 4 Weeks Post Dose 3-Pneumosil vs 4 Weeks Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 19, analysis 1]; OPA GMT Ratio-Type 7F = 3.89, 95% CI 2-sided [2.92 to 5.18]
Statistical Analysis 6: Comparison: 4 Weeks Post Dose 3-Pneumosil vs 4 Weeks Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 19, analysis 1]; OPA GMT Ratio-Type 9V = 6.85, 95% CI 2-sided [4.45 to 10.52]
Statistical Analysis 7: Comparison: 4 Weeks Post Dose 3-Pneumosil vs 4 Weeks Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 19, analysis 1]; OPA GMT Ratio-Type 14 = 2.45, 95% CI 2-sided [1.64 to 3.65]
Statistical Analysis 8: Comparison: 4 Weeks Post Dose 3-Pneumosil vs 4 Weeks Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 19, analysis 1]; OPA GMT Ratio-Type 19A = 3.64, 95% CI 2-sided [2.47 to 5.36]
Statistical Analysis 9: Comparison: 4 Weeks Post Dose 3-Pneumosil vs 4 Weeks Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 19, analysis 1]; OPA GMT Ratio-Type 19F = 2.38, 95% CI 2-sided [1.80 to 3.14]
Statistical Analysis 10: Comparison: 4 Weeks Post Dose 3-Pneumosil vs 4 Weeks Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 19, analysis 1]; OPA GMT Ratio-Type 23F = 4.97, 95% CI 2-sided [3.49 to 7.06]
Statistical Analysis 11: Comparison: 4 Weeks Post Dose 3-Synflorix vs 4 Weeks Post Booster-Synflorix; Test type: Other — [test comment as in outcome 19, analysis 1]; OPA GMT Ratio-Type 1 = 6.29, 95% CI 2-sided [4.97 to 7.96]
Statistical Analysis 12: Comparison: 4 Weeks Post Dose 3-Synflorix vs 4 Weeks Post Booster-Synflorix; Test type: Other — [test comment as in outcome 19, analysis 1]; OPA GMT Ratio-Type 5 = 3.19, 95% CI 2-sided [2.56 to 3.98]
Statistical Analysis 13: Comparison: 4 Weeks Post Dose 3-Synflorix vs 4 Weeks Post Booster-Synflorix; Test type: Other — [test comment as in outcome 19, analysis 1]; OPA GMT Ratio-Type 6A = 6.21, 95% CI 2-sided [3.55 to 10.84]
Statistical Analysis 14: Comparison: 4 Weeks Post Dose 3-Synflorix vs 4 Weeks Post Booster-Synflorix; Test type: Other — [test comment as in outcome 19, analysis 1]; OPA GMT Ratio-Type 6B = 3.25, 95% CI 2-sided [2.25 to 4.70]
Statistical Analysis 15: Comparison: 4 Weeks Post Dose 3-Synflorix vs 4 Weeks Post Booster-Synflorix; Test type: Other — [test comment as in outcome 19, analysis 1]; OPA GMT Ratio-Type 7F = 2.81, 95% CI 2-sided [2.13 to 3.69]
Statistical Analysis 16: Comparison: 4 Weeks Post Dose 3-Synflorix vs 4 Weeks Post Booster-Synflorix; Test type: Other — [test comment as in outcome 19, analysis 1]; OPA GMT Ratio-Type 9V = 2.95, 95% CI 2-sided [2.15 to 4.04]
Statistical Analysis 17: Comparison: 4 Weeks Post Dose 3-Synflorix vs 4 Weeks Post Booster-Synflorix; Test type: Other — [test comment as in outcome 19, analysis 1]; OPA GMT Ratio-Type 14 = 1.62, 95% CI 2-sided [1.06 to 2.46]
Statistical Analysis 18: Comparison: 4 Weeks Post Dose 3-Synflorix vs 4 Weeks Post Booster-Synflorix; Test type: Other — [test comment as in outcome 19, analysis 1]; OPA GMT Ratio-Type 19A = 5.98, 95% CI 2-sided [3.88 to 9.21]
Statistical Analysis 19: Comparison: 4 Weeks Post Dose 3-Synflorix vs 4 Weeks Post Booster-Synflorix; Test type: Other — [test comment as in outcome 19, analysis 1]; OPA GMT Ratio-Type 19F = 1.97, 95% CI 2-sided [1.45 to 2.68]
Statistical Analysis 20: Comparison: 4 Weeks Post Dose 3-Synflorix vs 4 Weeks Post Booster-Synflorix; Test type: Other — [test comment as in outcome 19, analysis 1]; OPA GMT Ratio-Type 23F = 5.73, 95% CI 2-sided [3.80 to 8.63]

20. Secondary Outcome: Serotype-specific OPA GMT and Treatment-Group GMT Ratios 4 Weeks After a Booster Dose
Description: Comparison of Serotype-specific booster responses (functional response) to PNEUMOSIL in comparison to Synflorix 4 weeks after a booster dose
Time Frame: 4 weeks post booster vaccination
Population: In a subset of subjects who got 3 primary series and a booster dose of study vaccines, had postdose immunogenicity measurement(s) with no major protocol deviations, serotype-specific OPA GMT and treatment group ratios of OPA GMT (with corresponding 95% CIs) were evaluated. Pooled PNEUMOSIL data was used for this analysis as per SAP
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Pneumosil | Synflorix
Number analyzed (Participants) | 99 | 100
titer
  OPA Type 1: number analyzed (Participants) | 98 | 97
  OPA Type 1 | 344.53 [261.77 to 453.46] | 187.16 [141.59 to 247.40]
  OPA Type 5 | 409.87 [312.35 to 537.84] | 360.59 [281.89 to 461.25]
  OPA Type 6A: number analyzed (Participants) | 98 | 95
  OPA Type 6A | 3063.37 [2328.56 to 4030.06] | 44.98 [25.86 to 78.25]
  OPA Type 6B: number analyzed (Participants) | 98 | 100
  OPA Type 6B | 2824.56 [2207.88 to 3613.50] | 1610.81 [1276.29 to 2033.01]
  OPA Type 7F | 6977.27 [5601.56 to 8690.85] | 4036.08 [3270.20 to 4981.32]
  OPA Type 9V: number analyzed (Participants) | 98 | 100
  OPA Type 9V | 1137.28 [862.30 to 1499.94] | 1229.05 [979.30 to 1542.50]
  OPA Type 14: number analyzed (Participants) | 97 | 99
  OPA Type 14 | 3114.71 [2331.38 to 4161.22] | 1411.94 [978.24 to 2037.92]
  OPA Type 19A: number analyzed (Participants) | 97 | 95
  OPA Type 19A | 645.56 [489.69 to 851.04] | 51.47 [32.40 to 81.76]
  OPA Type 19F: number analyzed (Participants) | 99 | 98
  OPA Type 19F | 1592.40 [1255.72 to 2019.35] | 1580.46 [1189.81 to 2099.38]
  OPA Type 23F | 3846.82 [2962.23 to 4995.58] | 1226.89 [967.91 to 1555.18]
Statistical Analysis 1: Comparison: Pneumosil vs Synflorix; Test type: Other — The vaccines will be compared using the ratios of the GMT ratios for the two treatment groups, i.e., the PNEUMOSIL ratio divided by the Synflorix ratio, and the corresponding 95% CIs based on log linear random effects models; OPA GMT Ratio-Type 1 = 1.84, 95% CI 2-sided [1.25 to 2.72]
Statistical Analysis 2: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 20, analysis 1]; OPA GMT Ratio-Type 5 = 1.14, 95% CI 2-sided [0.79 to 1.64]
Statistical Analysis 3: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 20, analysis 1]; OPA GMT Ratio-Type 6A = 68.10, 95% CI 2-sided [37.07 to 125.09]
Statistical Analysis 4: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 20, analysis 1]; OPA GMT Ratio-Type 6B = 1.75, 95% CI 2-sided [1.25 to 2.46]
Statistical Analysis 5: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 20, analysis 1]; OPA GMT Ratio-Type 7F = 1.73, 95% CI 2-sided [1.28 to 2.34]
Statistical Analysis 6: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 20, analysis 1]; OPA GMT Ratio-Type 9V = 0.93, 95% CI 2-sided [0.65 to 1.32]
Statistical Analysis 7: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 20, analysis 1]; OPA GMT Ratio-Type 14 = 2.21, 95% CI 2-sided [1.38 to 3.51]
Statistical Analysis 8: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 20, analysis 1]; OPA GMT Ratio-Type 19A = 12.54, 95% CI 2-sided [7.36 to 21.37]
Statistical Analysis 9: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 20, analysis 1]; OPA GMT Ratio-Type 19F = 1.01, 95% CI 2-sided [0.70 to 1.46]
Statistical Analysis 10: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 20, analysis 1]; OPA GMT Ratio-Type 23F = 3.14, 95% CI 2-sided [2.21 to 4.45]

21. Secondary Outcome: Number and Percentage of Subjects With EPI Vaccine Immune Responses (Measles, Rubella and Yellow Fever)
Description: Anti-measles IgG, anti-rubella IgG and anti-yellow fever neutralizing antibody titer
Time Frame: 4 weeks post booster vaccination
Population: Evaluated in a subset who got 3 primary doses and a booster dose, had postdose immunogenicity data with no major protocol deviations. Non-inferiority shown if 2-sided 95% CI for difference in response proportions (PNEUMOSIL-Synflorix) had lower limit >-0.10. For this, pooled PNUEMOSIL data was used as specified in SAP.
Measure: Count of Participants; unit: Participants
Groups:
- Pneumosil: Three primary doses + 1 booster dose of Pneumosil
- Synflorix: Three primary doses + 1 booster dose of Synflorix
Arm/Group | Pneumosil | Synflorix
Number analyzed (Participants) | 425 | 208
Participants
  Anti-Measles IgG ≥ 150 mIU/mL | 381 | 183
  Anti- Rubella IgG ≥ 4 IU/mL | 421 | 204
  Anti-Yellow Fever neutralizing Ab titer ≥ 1:8: number analyzed (Participants) | 424 | 208
  Anti-Yellow Fever neutralizing Ab titer ≥ 1:8 | 420 | 201
Statistical Analysis 1: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — Non-inferiority will be shown if a two-sided 95% CI for the treatment-group difference in response proportions (proportion with Synflorix co-administration minus proportion with PNEUMOSIL co-administration) has an upper limit of < 0.10; Absolute difference for measles = 1.7, 95% CI 2-sided [-3.3 to 7.4]
Statistical Analysis 2: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — [test comment as in outcome 21, analysis 1]; Absolute difference for rubella = 1.0, 95% CI 2-sided [-0.9 to 4.0]
Statistical Analysis 3: Comparison: Pneumosil vs Synflorix; Test type: Non-Inferiority — [test comment as in outcome 21, analysis 1]; Absolute difference for yellow fever = 2.4, 95% CI 2-sided [0.2 to 5.9]

22. Other Pre Specified Outcome: Proportions and Treatment Group Difference in Proportions of IgG Responders 1 Year Post Booster
Description: Treatment group proportions and treatment-group difference in proportions of IgG responders (IgG concentration ≥ 0.35 μg/mL)
Time Frame: One Year Post Booster Vaccination
Population: In a subset of subjects who got 3 primary and a booster dose of study vaccines, had postdose immunogenicity measurement(s) one year post booster with no major protocol deviations, serotype-specific IgG responders and treatment group comparisons (with corresponding 95% CIs) were evaluated. Pooled PNEUMOSIL data was used for this analysis as per SAP
Measure: Count of Participants; unit: Participants
Arm/Group | Pneumosil | Synflorix
Number analyzed (Participants) | 378 | 190
Participants
  Pn IgG Type 1: number analyzed (Participants) | 378 | 187
  Pn IgG Type 1 | 150 | 44
  Pn IgG Type 5: number analyzed (Participants) | 376 | 190
  Pn IgG Type 5 | 223 | 99
  Pn IgG Type 6A: number analyzed (Participants) | 375 | 188
  Pn IgG Type 6A | 306 | 97
  Pn IgG Type 6B: number analyzed (Participants) | 375 | 190
  Pn IgG Type 6B | 344 | 143
  Pn IgG Type 7F: number analyzed (Participants) | 378 | 189
  Pn IgG Type 7F | 296 | 117
  Pn IgG Type 9V: number analyzed (Participants) | 376 | 190
  Pn IgG Type 9V | 209 | 106
  Pn IgG Type 14 | 322 | 134
  Pn IgG Type 19A: number analyzed (Participants) | 375 | 184
  Pn IgG Type 19A | 316 | 128
  Pn IgG Type 19F: number analyzed (Participants) | 377 | 186
  Pn IgG Type 19F | 301 | 174
  Pn IgG Type 23F: number analyzed (Participants) | 377 | 186
  Pn IgG Type 23F | 224 | 79
Statistical Analysis 1: Comparison: Pneumosil vs Synflorix; Test type: Other — Treatment group difference in proportions; Absolute Difference for Type 1 = 16.2, 95% CI 2-sided [8.0 to 23.7]
Statistical Analysis 2: Comparison: Pneumosil vs Synflorix; Test type: Other — Treatment group difference in proportions; Absolute Difference for Type 5 = 7.2, 95% CI 2-sided [-1.4 to 15.8]
Statistical Analysis 3: Comparison: Pneumosil vs Synflorix; Test type: Other — Treatment group difference in proportions; Absolute Difference for Type 6A = 30.0, 95% CI 2-sided [21.8 to 38.1]
Statistical Analysis 4: Comparison: Pneumosil vs Synflorix; Test type: Other — Treatment group difference in proportions; Absolute Difference for Type 6B = 16.5, 95% CI 2-sided [10.1 to 23.6]
Statistical Analysis 5: Comparison: Pneumosil vs Synflorix; Test type: Other — Treatment group difference in proportions; Absolute Difference for Type 7F = 16.4, 95% CI 2-sided [8.4 to 24.5]
Statistical Analysis 6: Comparison: Pneumosil vs Synflorix; Test type: Other — Treatment group difference in proportions; Absolute Difference for Type 9V = -0.2, 95% CI 2-sided [-8.8 to 8.5]
Statistical Analysis 7: Comparison: Pneumosil vs Synflorix; Test type: Other — Treatment group difference in proportions; Absolute Difference for Type 14 = 14.7, 95% CI 2-sided [7.5 to 22.3]
Statistical Analysis 8: Comparison: Pneumosil vs Synflorix; Test type: Other — Treatment group difference in proportions; Absolute Difference for Type 19A = 14.7, 95% CI 2-sided [7.3 to 22.5]
Statistical Analysis 9: Comparison: Pneumosil vs Synflorix; Test type: Other — Treatment group difference in proportions; Absolute Difference for Type 19F = -13.7, 95% CI 2-sided [-19.0 to -8.0]
Statistical Analysis 10: Comparison: Pneumosil vs Synflorix; Test type: Other — Treatment group difference in proportions; Absolute Difference for Type 23F = 16.9, 95% CI 2-sided [8.2 to 25.4]

23. Other Pre Specified Outcome: Serotype-specific Geometric Mean Concentration of IgG Antibody Response and Treatment-Group GMC Ratios One Year Post Booster
Description: Comparison of Serotype-specific immune persistence responses (antibody concentrations) to PNEUMOSIL in comparison to Synflorix one year post booster
Time Frame: One year post booster vaccination
Population: Subset of subjects who got 3 primary and a booster dose of study vaccines, had postdose immunogenicity measurement(s) one year post booster with no major protocol deviations, serotype-specific GMC of IgG Antibody and treatment group ratios of IgG GMCs (with corresponding 95% CIs) evaluated. Pooled PNEUMOSIL data was used for this analysis
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Pneumosil | Synflorix
Number analyzed (Participants) | 378 | 190
µg/mL
  Pn IgG Type 1: number analyzed (Participants) | 378 | 187
  Pn IgG Type 1 | 0.30 [0.28 to 0.32] | 0.18 [0.16 to 0.21]
  Pn IgG Type 5: number analyzed (Participants) | 376 | 190
  Pn IgG Type 5 | 0.40 [0.37 to 0.44] | 0.34 [0.29 to 0.39]
  Pn IgG Type 6A: number analyzed (Participants) | 375 | 188
  Pn IgG Type 6A | 0.73 [0.67 to 0.80] | 0.31 [0.26 to 0.36]
  Pn IgG Type 6B: number analyzed (Participants) | 375 | 190
  Pn IgG Type 6B | 0.90 [0.84 to 0.97] | 0.62 [0.55 to 0.71]
  Pn IgG Type 7F: number analyzed (Participants) | 378 | 189
  Pn IgG Type 7F | 0.64 [0.59 to 0.69] | 0.49 [0.44 to 0.55]
  Pn IgG Type 9V: number analyzed (Participants) | 376 | 190
  Pn IgG Type 9V | 0.38 [0.35 to 0.42] | 0.41 [0.36 to 0.46]
  Pn IgG Type 14 | 0.99 [0.89 to 1.10] | 0.71 [0.59 to 0.85]
  Pn IgG Type 19A: number analyzed (Participants) | 375 | 184
  Pn IgG Type 19A | 0.91 [0.81 to 1.01] | 0.66 [0.55 to 0.78]
  Pn IgG Type 19F: number analyzed (Participants) | 377 | 186
  Pn IgG Type 19F | 0.82 [0.73 to 0.92] | 1.35 [1.17 to 1.55]
  Pn IgG Type 23F: number analyzed (Participants) | 377 | 186
  Pn IgG Type 23F | 0.43 [0.39 to 0.48] | 0.29 [0.25 to 0.34]
Statistical Analysis 1: Comparison: Pneumosil vs Synflorix; Test type: Other — The vaccines were compared using the ratios of the GMC ratios for the two treatment groups, i.e., the PNEUMOSIL ratio divided by the Synflorix ratio, and the corresponding 95% CIs; Pn IgG type 1 GMC Ratio = 1.64, 95% CI 2-sided [1.42 to 1.89]
Statistical Analysis 2: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 23, analysis 1]; Pn IgG type 5 GMC Ratio = 1.20, 95% CI 2-sided [1.03 to 1.40]
Statistical Analysis 3: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 23, analysis 1]; Pn IgG type 6A GMC Ratio = 2.36, 95% CI 2-sided [2.01 to 2.78]
Statistical Analysis 4: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 23, analysis 1]; Pn IgG type 6B GMC Ratio = 1.45, 95% CI 2-sided [1.27 to 1.66]
Statistical Analysis 5: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 23, analysis 1]; Pn IgG type 7F GMC Ratio = 1.29, 95% CI 2-sided [1.12 to 1.49]
Statistical Analysis 6: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 23, analysis 1]; Pn IgG type 9V GMC Ratio = 0.94, 95% CI 2-sided [0.81 to 1.09]
Statistical Analysis 7: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 23, analysis 1]; Pn IgG type 14 GMC Ratio = 1.41, 95% CI 2-sided [1.15 to 1.72]
Statistical Analysis 8: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 23, analysis 1]; Pn IgG type 19A GMC Ratio = 1.38, 95% CI 2-sided [1.14 to 1.68]
Statistical Analysis 9: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 23, analysis 1]; Pn IgG type 19F GMC Ratio = 0.61, 95% CI 2-sided [0.50 to 0.74]
Statistical Analysis 10: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 23, analysis 1]; Pn IgG type 23F GMC Ratio = 1.50, 95% CI 2-sided [1.24 to 1.81]

24. Other Pre Specified Outcome: Comparison of Serotype-specific Geometric Mean Concentration of IgG Antibody Response 4 Weeks After a Booster Dose to One Year After a Booster Dose
Description: Comparison of Serotype-specific responses (antibody concentrations) measured by ELISA from 4 weeks after a booster dose to one year after a booster dose
Time Frame: One year post booster vaccination
Population: Subset who got 3 primary series+booster dose of study vaccines, had postdose immunogenicity measurements post booster, no major PDs, comparisons based on ratios of IgG GMC one year post booster to IgG GMC four weeks post booster. Comparison done using ratios of the ratios for the 2 treatment groups & corresponding 95% CIs.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Groups:
- 4 Weeks Post Booster Dose-Pneumosil; One Year Post Booster-Pneumosil: Three doses + 1 booster dose of Pneumosil in a subset
- 4 Weeks Post Booster Dose-Synflorix; One Year Post Booster-Synflorix: Three doses + 1 booster dose of Synflorix in a subset
Arm/Group | 4 Weeks Post Booster Dose-Pneumosil | One Year Post Booster-Pneumosil | 4 Weeks Post Booster Dose-Synflorix | One Year Post Booster-Synflorix
Number analyzed (Participants) | 378 | 378 | 189 | 190
µg/mL
  Pn IgG Type 1: number analyzed (Participants) | 378 | 378 | 189 | 187
  Pn IgG Type 1 | 5.87 [5.36 to 6.42] | 0.30 [0.28 to 0.32] | 2.52 [2.21 to 2.88] | 0.18 [0.16 to 0.21]
  Pn IgG Type 5: number analyzed (Participants) | 378 | 376 | 188 | 190
  Pn IgG Type 5 | 1.35 [1.24 to 1.46] | 0.40 [0.37 to 0.44] | 0.85 [0.77 to 0.95] | 0.34 [0.29 to 0.39]
  Pn IgG Type 6A: number analyzed (Participants) | 377 | 375 | 189 | 188
  Pn IgG Type 6A | 4.86 [4.37 to 5.41] | 0.73 [0.67 to 0.80] | 0.43 [0.36 to 0.51] | 0.31 [0.26 to 0.36]
  Pn IgG Type 6B: number analyzed (Participants) | 376 | 375 | 189 | 190
  Pn IgG Type 6B | 8.48 [7.84 to 9.18] | 0.90 [0.84 to 0.97] | 4.45 [3.99 to 4.97] | 0.62 [0.55 to 0.71]
  Pn IgG Type 7F: number analyzed (Participants) | 378 | 378 | 189 | 189
  Pn IgG Type 7F | 6.40 [5.87 to 6.97] | 0.64 [0.59 to 0.69] | 4.14 [3.72 to 4.60] | 0.49 [0.44 to 0.55]
  Pn IgG Type 9V: number analyzed (Participants) | 377 | 376 | 189 | 190
  Pn IgG Type 9V | 1.86 [1.72 to 2.01] | 0.38 [0.35 to 0.42] | 2.08 [1.87 to 2.32] | 0.41 [0.36 to 0.46]
  Pn IgG Type 14: number analyzed (Participants) | 374 | 378 | 184 | 190
  Pn IgG Type 14 | 6.58 [5.80 to 7.46] | 0.99 [0.89 to 1.10] | 4.61 [3.83 to 5.56] | 0.71 [0.59 to 0.85]
  Pn IgG Type 19A: number analyzed (Participants) | 376 | 375 | 185 | 184
  Pn IgG Type 19A | 4.02 [3.66 to 4.42] | 0.91 [0.81 to 1.01] | 1.00 [0.82 to 1.22] | 0.66 [0.55 to 0.78]
  Pn IgG Type 19F: number analyzed (Participants) | 371 | 377 | 185 | 186
  Pn IgG Type 19F | 6.17 [5.65 to 6.73] | 0.82 [0.73 to 0.92] | 9.80 [8.72 to 11.02] | 1.35 [1.17 to 1.55]
  Pn IgG Type 23F: number analyzed (Participants) | 378 | 377 | 189 | 186
  Pn IgG Type 23F | 4.03 [3.66 to 4.45] | 0.43 [0.39 to 0.48] | 2.12 [1.86 to 2.42] | 0.29 [0.25 to 0.34]
Statistical Analysis 1: Comparison: 4 Weeks Post Booster Dose-Pneumosil vs One Year Post Booster-Pneumosil; Test type: Other — The comparisons were based on the ratio of IgG GMC one year post-booster to the IgG GMC 4 weeks post booster in the Booster Cohort; Pn IgG type 1 GMC Ratio = 0.05, 95% CI 2-sided [0.05 to 0.06]
Statistical Analysis 2: Comparison: 4 Weeks Post Booster Dose-Pneumosil vs One Year Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 24, analysis 1]; Pn IgG type 5 GMC Ratio = 0.30, 95% CI 2-sided [0.27 to 0.33]
Statistical Analysis 3: Comparison: 4 Weeks Post Booster Dose-Pneumosil vs One Year Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 24, analysis 1]; Pn IgG type 6A GMC Ratio = 0.15, 95% CI 2-sided [0.13 to 0.16]
Statistical Analysis 4: Comparison: 4 Weeks Post Booster Dose-Pneumosil vs One Year Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 24, analysis 1]; Pn IgG type 6B GMC Ratio = 0.11, 95% CI 2-sided [0.10 to 0.11]
Statistical Analysis 5: Comparison: 4 Weeks Post Booster Dose-Pneumosil vs One Year Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 24, analysis 1]; Pn IgG type 7F GMC Ratio = 0.10, 95% CI 2-sided [0.09 to 0.11]
Statistical Analysis 6: Comparison: 4 Weeks Post Booster Dose-Pneumosil vs One Year Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 24, analysis 1]; Pn IgG type 9V GMC Ratio = 0.21, 95% CI 2-sided [0.19 to 0.23]
Statistical Analysis 7: Comparison: 4 Weeks Post Booster Dose-Pneumosil vs One Year Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 24, analysis 1]; Pn IgG type 14 GMC Ratio = 0.15, 95% CI 2-sided [0.13 to 0.17]
Statistical Analysis 8: Comparison: 4 Weeks Post Booster Dose-Pneumosil vs One Year Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 24, analysis 1]; Pn IgG type 19A GMC Ratio = 0.23, 95% CI 2-sided [0.20 to 0.26]
Statistical Analysis 9: Comparison: 4 Weeks Post Booster Dose-Pneumosil vs One Year Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 24, analysis 1]; Pn IgG type 19F GMC Ratio = 0.14, 95% CI 2-sided [0.12 to 0.15]
Statistical Analysis 10: Comparison: 4 Weeks Post Booster Dose-Pneumosil vs One Year Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 24, analysis 1]; Pn IgG type 23F GMC Ratio = 0.11, 95% CI 2-sided [0.10 to 0.12]
Statistical Analysis 11: Comparison: 4 Weeks Post Booster Dose-Synflorix vs One Year Post Booster-Synflorix; Test type: Other — [test comment as in outcome 24, analysis 1]; Pn IgG type 1 GMC Ratio = 0.07, 95% CI 2-sided [0.06 to 0.08]
Statistical Analysis 12: Comparison: 4 Weeks Post Booster Dose-Synflorix vs One Year Post Booster-Synflorix; Test type: Other — [test comment as in outcome 24, analysis 1]; Pn IgG type 5 GMC Ratio = 0.40, 95% CI 2-sided [0.35 to 0.45]
Statistical Analysis 13: Comparison: 4 Weeks Post Booster Dose-Synflorix vs One Year Post Booster-Synflorix; Test type: Other — [test comment as in outcome 24, analysis 1]; Pn IgG type 6A GMC Ratio = 0.73, 95% CI 2-sided [0.62 to 0.86]
Statistical Analysis 14: Comparison: 4 Weeks Post Booster Dose-Synflorix vs One Year Post Booster-Synflorix; Test type: Other — [test comment as in outcome 24, analysis 1]; Pn IgG type 6B GMC Ratio = 0.14, 95% CI 2-sided [0.12 to 0.16]
Statistical Analysis 15: Comparison: 4 Weeks Post Booster Dose-Synflorix vs One Year Post Booster-Synflorix; Test type: Other — [test comment as in outcome 24, analysis 1]; Pn IgG type 7F GMC Ratio = 0.12, 95% CI 2-sided [0.11 to 0.13]
Statistical Analysis 16: Comparison: 4 Weeks Post Booster Dose-Synflorix vs One Year Post Booster-Synflorix; Test type: Other — [test comment as in outcome 24, analysis 1]; Pn IgG type 9V GMC Ratio = 0.20, 95% CI 2-sided [0.18 to 0.22]
Statistical Analysis 17: Comparison: 4 Weeks Post Booster Dose-Synflorix vs One Year Post Booster-Synflorix; Test type: Other — [test comment as in outcome 24, analysis 1]; Pn IgG type 14 GMC Ratio = 0.15, 95% CI 2-sided [0.13 to 0.19]
Statistical Analysis 18: Comparison: 4 Weeks Post Booster Dose-Synflorix vs One Year Post Booster-Synflorix; Test type: Other — [test comment as in outcome 24, analysis 1]; Pn IgG type 19A GMC Ratio = 0.64, 95% CI 2-sided [0.52 to 0.78]
Statistical Analysis 19: Comparison: 4 Weeks Post Booster Dose-Synflorix vs One Year Post Booster-Synflorix; Test type: Other — [test comment as in outcome 24, analysis 1]; Pn IgG type 19F GMC Ratio = 0.14, 95% CI 2-sided [0.12 to 0.16]
Statistical Analysis 20: Comparison: 4 Weeks Post Booster Dose-Synflorix vs One Year Post Booster-Synflorix; Test type: Other — [test comment as in outcome 24, analysis 1]; Pn IgG type 23F GMC Ratio = 0.14, 95% CI 2-sided [0.12 to 0.16]

25. Other Pre Specified Outcome: Treatment Group Proportions and Treatment-group Difference in Proportions of Functional Antibody Responders (OPA) One Year Post Booster
Description: Serotype-specific functional antibody titer measured by OPA
Time Frame: One year post booster vaccination
Population: Subset of subjects who got 3 primary doses + booster dose, had postdose immunogenicity measurement one year after booster, no major protocol deviations, functional immune responses induced by PNEUMOSIL were compared to Synflorix for 10 serotypes OPA Type 1[OPA seroresponse rate (titer≥1:8)] differences.Pooled PNEUMOSIL data was used.
Measure: Count of Participants; unit: Participants
Arm/Group | Pneumosil | Synflorix
Number analyzed (Participants) | 50 | 50
Participants
  OPA Type 1: number analyzed (Participants) | 50 | 47
  OPA Type 1 | 27 | 14
  OPA Type 5: number analyzed (Participants) | 44 | 47
  OPA Type 5 | 39 | 37
  OPA Type 6A: number analyzed (Participants) | 50 | 49
  OPA Type 6A | 42 | 9
  OPA Type 6B: number analyzed (Participants) | 49 | 48
  OPA Type 6B | 43 | 31
  OPA Type 7F: number analyzed (Participants) | 50 | 49
  OPA Type 7F | 50 | 48
  OPA Type 9V: number analyzed (Participants) | 43 | 40
  OPA Type 9V | 43 | 40
  OPA Type 14: number analyzed (Participants) | 49 | 47
  OPA Type 14 | 45 | 41
  OPA Type 19A: number analyzed (Participants) | 49 | 45
  OPA Type 19A | 43 | 24
  OPA Type 19F: number analyzed (Participants) | 48 | 45
  OPA Type 19F | 44 | 39
  OPA Type 23F: number analyzed (Participants) | 49 | 43
  OPA Type 23F | 49 | 43
Statistical Analysis 1: Comparison: Pneumosil vs Synflorix; Test type: Other — Serotype specific functional antibody responses measured by OPA titer to Pneumosil in comparison with Synflorix for each of the 10 serotypes one year post booster; OPA Type 1 = 24.2, 95% CI 2-sided [4.5 to 42.1]
Statistical Analysis 2: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 25, analysis 1]; OPA Type 5 = 9.9, 95% CI 2-sided [-5.8 to 25.5]
Statistical Analysis 3: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 25, analysis 1]; OPA Type 6A = 65.6, 95% CI 2-sided [48.3 to 78.0]
Statistical Analysis 4: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 25, analysis 1]; OPA Type 6B = 23.2, 95% CI 2-sided [6.4 to 39.4]
Statistical Analysis 5: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 25, analysis 1]; OPA Type 7F = 2.0, 95% CI 2-sided [-5.2 to 10.8]
Statistical Analysis 6: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 25, analysis 1]; OPA Type 9V = 0.0 — CI could not be computed due to 100% response rate
Statistical Analysis 7: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 25, analysis 1]; OPA Type14 = 4.6, 95% CI 2-sided [-8.5 to 18.3]
Statistical Analysis 8: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 25, analysis 1]; OPA Type 19A = 34.4, 95% CI 2-sided [16.5 to 50.8]
Statistical Analysis 9: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 25, analysis 1]; OPA Type 19F = 5.0, 95% CI 2-sided [-8.4 to 19.2]
Statistical Analysis 10: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 25, analysis 1]; OPA Type 23F = 0.0 — CI could not be computed due to 100% response rate

26. Other Pre Specified Outcome: Serotype-specific OPA Geometric Mean Titer One Year Post Booster
Description: Serotype-specific functional antibody titer measured by OPA and expressed as OPA GMT in a subset one year post booster
Time Frame: One year post booster vaccination
Population: In a subset of subjects who got 3 primary + booster dose of study vaccines, had postdose immunogenicity measurement one year post booster and no major protocol deviations, functional immune responses induced by PNEUMOSIL were compared to Synflorix for 10 serotypes, i.e., ratio of OPA GMTs (and corresponding 95% CIs).Pooled PNEUMOSIL data was used.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Pneumosil | Synflorix
Number analyzed (Participants) | 50 | 50
Titer
  OPA Type 1: number analyzed (Participants) | 50 | 47
  OPA Type 1 | 11.0 [8.0 to 15.1] | 8.7 [5.9 to 12.9]
  OPA Type 5: number analyzed (Participants) | 44 | 47
  OPA Type 5 | 41.4 [27.6 to 62.0] | 31.6 [20.0 to 50.1]
  OPA Type 6A: number analyzed (Participants) | 50 | 49
  OPA Type 6A | 118.1 [61.6 to 226.5] | 8.3 [5.0 to 13.6]
  OPA Type 6B: number analyzed (Participants) | 49 | 48
  OPA Type 6B | 116.3 [74.9 to 180.6] | 31.1 [20.5 to 47.2]
  OPA Type 7F: number analyzed (Participants) | 50 | 49
  OPA Type 7F | 1765.9 [1238.1 to 2518.8] | 1851.8 [1251.3 to 2740.5]
  OPA Type 9V: number analyzed (Participants) | 43 | 40
  OPA Type 9V | 114.5 [63.8 to 205.5] | 158.2 [86.3 to 289.9]
  OPA Type 14: number analyzed (Participants) | 49 | 47
  OPA Type 14 | 215.1 [126.2 to 366.6] | 193.4 [107.9 to 346.6]
  OPA Type 19A: number analyzed (Participants) | 49 | 45
  OPA Type 19A | 89.7 [50.2 to 160.3] | 17.6 [11.0 to 28.3]
  OPA Type 19F: number analyzed (Participants) | 48 | 45
  OPA Type 19F | 133.5 [68.2 to 261.1] | 139.8 [78.3 to 249.8]
  OPA Type 23F: number analyzed (Participants) | 49 | 43
  OPA Type 23F | 393.8 [219.3 to 707.4] | 91.6 [54.0 to 155.3]
Statistical Analysis 1: Comparison: Pneumosil vs Synflorix; Test type: Other — Serotype specific functional antibody responses measured by OPA to Pneumosil in comparison with Synflorix for each of the 10 serotypes (GMT Ratio) one year post booster dose; OPA GMT Ratio-Type 1 = 1.3, 95% CI 2-sided [0.8 to 2.1]
Statistical Analysis 2: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 26, analysis 1]; OPA GMT Ratio-Type 5 = 1.3, 95% CI 2-sided [0.7 to 2.4]
Statistical Analysis 3: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 26, analysis 1]; OPA GMT Ratio-Type 6A = 14.3, 95% CI 2-sided [6.3 to 32.1]
Statistical Analysis 4: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 26, analysis 1]; OPA GMT Ratio-Type 6B = 3.7, 95% CI 2-sided [2.1 to 6.8]
Statistical Analysis 5: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 26, analysis 1]; OPA GMT Ratio-Type 7F = 1.0, 95% CI 2-sided [0.6 to 1.6]
Statistical Analysis 6: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 26, analysis 1]; OPA GMT Ratio-Type 9V = 0.7, 95% CI 2-sided [0.3 to 1.7]
Statistical Analysis 7: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 26, analysis 1]; OPA GMT Ratio-Type 14 = 1.1, 95% CI 2-sided [0.5 to 2.4]
Statistical Analysis 8: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 26, analysis 1]; OPA GMT Ratio-Type 19A = 5.1, 95% CI 2-sided [2.4 to 10.8]
Statistical Analysis 9: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 26, analysis 1]; OPA GMT Ratio-Type 19F = 1.0, 95% CI 2-sided [0.4 to 2.3]
Statistical Analysis 10: Comparison: Pneumosil vs Synflorix; Test type: Other — [test comment as in outcome 26, analysis 1]; OPA GMT Ratio-Type 23F = 4.3, 95% CI 2-sided [2.0 to 9.4]

27. Other Pre Specified Outcome: Comparison of Functional Response (OPA) From 4 Weeks After a Booster Dose to One Year Post Booster Dose
Description: Comparison of Serotype-specific booster responses (functional response-OPA) from 4 weeks after a booster dose to one year post booster
Time Frame: One year post booster vaccination
Population: In a subset who got 3 primary series+booster dose of study vaccines, had postdose immunogenicity measurements & no major PDs, comparisons based on ratios of OPA GMT one year post booster to OPA GMT 4 weeks post booster. Comparison done using ratios of the ratios for the 2 treatment groups (PNEUMOSIL ratio/Synflorix ratio), & corresponding 95% CIs.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | 4 Weeks Post Booster Dose-Pneumosil | One Year Post Booster-Pneumosil | 4 Weeks Post Booster Dose-Synflorix | One Year Post Booster-Synflorix
Number analyzed (Participants) | 88 | 50 | 91 | 50
Titer
  OPA Type 1: number analyzed (Participants) | 87 | 50 | 89 | 47
  OPA Type 1 | 345.8 [256.7 to 465.9] | 11.0 [8.0 to 15.1] | 191.7 [144.8 to 253.7] | 8.7 [5.9 to 12.9]
  OPA Type 5: number analyzed (Participants) | 88 | 44 | 91 | 47
  OPA Type 5 | 422.9 [315.4 to 567.1] | 41.4 [27.6 to 62.0] | 369.6 [289.0 to 472.8] | 31.6 [20.0 to 50.1]
  OPA Type 6A: number analyzed (Participants) | 87 | 50 | 87 | 49
  OPA Type 6A | 3119.4 [2313.3 to 4206.5] | 118.1 [61.6 to 226.5] | 49.9 [27.9 to 89.3] | 8.3 [5.0 to 13.6]
  OPA Type 6B: number analyzed (Participants) | 87 | 49 | 91 | 48
  OPA Type 6B | 3012.0 [2309.2 to 3928.6] | 116.3 [74.9 to 180.6] | 1613.8 [1258.1 to 2070.1] | 31.1 [20.5 to 47.2]
  OPA Type 7F: number analyzed (Participants) | 88 | 50 | 91 | 49
  OPA Type 7F | 6757.8 [5305.8 to 8607.2] | 1765.9 [1238.1 to 2518.8] | 4033.5 [3251.2 to 5004.1] | 1851.8 [1251.3 to 2740.5]
  OPA Type 9V: number analyzed (Participants) | 87 | 43 | 91 | 40
  OPA Type 9V | 1114.9 [828.6 to 1500.2] | 114.5 [63.8 to 205.5] | 1231.4 [966.5 to 1568.9] | 158.2 [86.3 to 289.9]
  OPA Type 14: number analyzed (Participants) | 87 | 49 | 90 | 47
  OPA Type 14 | 3128.9 [2279.9 to 4294.0] | 215.1 [126.2 to 366.6] | 1423.1 [962.7 to 2103.8] | 193.4 [107.9 to 346.6]
  OPA Type 19A: number analyzed (Participants) | 86 | 49 | 86 | 45
  OPA Type 19A | 643.6 [479.0 to 864.9] | 89.7 [50.2 to 160.3] | 54.6 [34.1 to 87.4] | 17.6 [11.0 to 28.3]
  OPA Type 19F: number analyzed (Participants) | 88 | 48 | 89 | 45
  OPA Type 19F | 1651.1 [1282.4 to 2125.8] | 133.5 [68.2 to 261.1] | 1611.8 [1227.5 to 2116.4] | 139.8 [78.3 to 249.8]
  OPA Type 23F: number analyzed (Participants) | 88 | 49 | 91 | 43
  OPA Type 23F | 3933.9 [2961.7 to 5225.1] | 393.8 [219.3 to 707.4] | 1219.8 [946.8 to 1571.5] | 91.6 [54.0 to 155.3]
Statistical Analysis 1: Comparison: 4 Weeks Post Booster Dose-Pneumosil vs One Year Post Booster-Pneumosil; Test type: Other — The comparisons were based on OPA GMTs 4 weeks post booster and one year post booster for the OPA subset of the booster cohort; OPA GMT Ratio-Type 1 = 0.04, 95% CI 2-sided [0.03 to 0.06]
Statistical Analysis 2: Comparison: 4 Weeks Post Booster Dose-Pneumosil vs One Year Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 27, analysis 1]; OPA GMT Ratio-Type 5 = 0.11, 95% CI 2-sided [0.09 to 0.14]
Statistical Analysis 3: Comparison: 4 Weeks Post Booster Dose-Pneumosil vs One Year Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 27, analysis 1]; OPA GMT Ratio-Type 6A = 0.05, 95% CI 2-sided [0.03 to 0.08]
Statistical Analysis 4: Comparison: 4 Weeks Post Booster Dose-Pneumosil vs One Year Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 27, analysis 1]; OPA GMT Ratio-Type 6B = 0.05, 95% CI 2-sided [0.03 to 0.07]
Statistical Analysis 5: Comparison: 4 Weeks Post Booster Dose-Pneumosil vs One Year Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 27, analysis 1]; OPA GMT Ratio-Type 7F = 0.26, 95% CI 2-sided [0.18 to 0.38]
Statistical Analysis 6: Comparison: 4 Weeks Post Booster Dose-Pneumosil vs One Year Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 27, analysis 1]; OPA GMT Ratio-Type 9V = 0.12, 95% CI 2-sided [0.06 to 0.23]
Statistical Analysis 7: Comparison: 4 Weeks Post Booster Dose-Pneumosil vs One Year Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 27, analysis 1]; OPA GMT Ratio-Type 14 = 0.07, 95% CI 2-sided [0.05 to 0.11]
Statistical Analysis 8: Comparison: 4 Weeks Post Booster Dose-Pneumosil vs One Year Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 27, analysis 1]; OPA GMT Ratio-Type 19A = 0.16, 95% CI 2-sided [0.09 to 0.30]
Statistical Analysis 9: Comparison: 4 Weeks Post Booster Dose-Pneumosil vs One Year Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 27, analysis 1]; OPA GMT Ratio-Type 19F = 0.09, 95% CI 2-sided [0.05 to 0.18]
Statistical Analysis 10: Comparison: 4 Weeks Post Booster Dose-Pneumosil vs One Year Post Booster-Pneumosil; Test type: Other — [test comment as in outcome 27, analysis 1]; OPA GMT Ratio-Type 23F = 0.12, 95% CI 2-sided [0.08 to 0.18]
Statistical Analysis 11: Comparison: 4 Weeks Post Booster Dose-Synflorix vs One Year Post Booster-Synflorix; Test type: Other — [test comment as in outcome 27, analysis 1]; OPA GMT Ratio-Type 1 = 0.04, 95% CI 2-sided [0.03 to 0.06]
Statistical Analysis 12: Comparison: 4 Weeks Post Booster Dose-Synflorix vs One Year Post Booster-Synflorix; Test type: Other — [test comment as in outcome 27, analysis 1]; OPA GMT Ratio-Type 5 = 0.07, 95% CI 2-sided [0.05 to 0.10]
Statistical Analysis 13: Comparison: 4 Weeks Post Booster Dose-Synflorix vs One Year Post Booster-Synflorix; Test type: Other — [test comment as in outcome 27, analysis 1]; OPA GMT Ratio-Type 6A = 0.21, 95% CI 2-sided [0.09 to 0.48]
Statistical Analysis 14: Comparison: 4 Weeks Post Booster Dose-Synflorix vs One Year Post Booster-Synflorix; Test type: Other — [test comment as in outcome 27, analysis 1]; OPA GMT Ratio-Type 6B = 0.02, 95% CI 2-sided [0.01 to 0.03]
Statistical Analysis 15: Comparison: 4 Weeks Post Booster Dose-Synflorix vs One Year Post Booster-Synflorix; Test type: Other — [test comment as in outcome 27, analysis 1]; OPA GMT Ratio-Type 7F = 0.44, 95% CI 2-sided [0.30 to 0.65]
Statistical Analysis 16: Comparison: 4 Weeks Post Booster Dose-Synflorix vs One Year Post Booster-Synflorix; Test type: Other — [test comment as in outcome 27, analysis 1]; OPA GMT Ratio-Type 9V = 0.11, 95% CI 2-sided [0.06 to 0.20]
Statistical Analysis 17: Comparison: 4 Weeks Post Booster Dose-Synflorix vs One Year Post Booster-Synflorix; Test type: Other — [test comment as in outcome 27, analysis 1]; OPA GMT Ratio-Type 14 = 0.11, 95% CI 2-sided [0.06 to 0.22]
Statistical Analysis 18: Comparison: 4 Weeks Post Booster Dose-Synflorix vs One Year Post Booster-Synflorix; Test type: Other — [test comment as in outcome 27, analysis 1]; OPA GMT Ratio-Type 19A = 0.26, 95% CI 2-sided [0.14 to 0.49]
Statistical Analysis 19: Comparison: 4 Weeks Post Booster Dose-Synflorix vs One Year Post Booster-Synflorix; Test type: Other — [test comment as in outcome 27, analysis 1]; OPA GMT Ratio-Type 19F = 0.09, 95% CI 2-sided [0.06 to 0.14]
Statistical Analysis 20: Comparison: 4 Weeks Post Booster Dose-Synflorix vs One Year Post Booster-Synflorix; Test type: Other — [test comment as in outcome 27, analysis 1]; OPA GMT Ratio-Type 23F = 0.07, 95% CI 2-sided [0.05 to 0.12]

ADVERSE EVENTS:
Time Frame: Recording and reporting of all AEs occurred from signing of the ICF (6-8 weeks of age) through the EOS visit for each subject enrolled in the priming phase of the study (upto 18-20 weeks of age), and through Visit 6 for each study subject enrolled in the booster phase (upto 12 months of age). Subjects included in the third phase for immune persistence evaluation, serious adverse events were monitored from 4 weeks post booster to 12 months after booster.
Description: Immediate solicited local and systemic reactogenicity events and vital signs were assessed 30 minutes following vaccination in all subjects. Half of the subjects in each treatment group were randomly selected to be part of the primary reactogenicity cohort. These subjects and those who received a booster dose were monitored daily at home for 6 days after each study vaccine dose by field workers. As stated in the SAP, pooled PNEUMOSIL data was used for safety analyses.
Groups:
- Pneumosil: Three doses of Pneumosil in primary series cohort and three + 1 booster dose in booster cohort
- Synflorix: Three doses of Synflorix in primary series cohort and three + 1 booster dose in booster cohort
Arm/Group | Pneumosil | Synflorix
All-Cause Mortality (participants affected / at risk) | 1/1503 | 2/747
Serious Adverse Events (participants affected / at risk) | 51/1503 | 26/747
Other Adverse Events (participants affected / at risk) | 1131/1503 | 572/747
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pneumosil (N=1503) | Synflorix (N=747)
Bronchiolitis (Infections and infestations) | 14 (14) | 4 (4)
Gastroenteritis (Infections and infestations) | 15 (17) | 9 (9)
Pneumonia (Infections and infestations) | 4 (4) | 6 (6)
Dysentery (Infections and infestations) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1)
HIV infection WHO clinical stage IV (Infections and infestations) | 0 (0) | 1 (1)
Meningitis pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Perinatal HIV infection (Infections and infestations) | 0 (0) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 3 (3) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0)
Fallot's tetralogy (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Trisomy 21 (Congenital, familial and genetic disorders) | 2 (2) | 0 (0)
Atrioventricular septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Developmental delay (General disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pneumosil (N=1503) | Synflorix (N=747)
Upper respiratory tract infection (Infections and infestations) | 730 (1041) | 379 (552)
Furuncle (Infections and infestations) | 150 (183) | 65 (77)
Gastroenteritis (Infections and infestations) | 154 (169) | 76 (80)
Conjunctivitis (Infections and infestations) | 110 (116) | 64 (67)
Bronchiolitis (Infections and infestations) | 59 (65) | 42 (47)
Tinea infection (Infections and infestations) | 62 (62) | 22 (22)
Febrile infection (Infections and infestations) | 52 (54) | 25 (28)
Pneumonia (Infections and infestations) | 41 (44) | 21 (21)
Tinea capitis (Infections and infestations) | 29 (30) | 22 (23)
Oral candidiasis (Infections and infestations) | 33 (37) | 15 (15)
Body tinea (Infections and infestations) | 29 (29) | 18 (18)
Impetigo (Infections and infestations) | 27 (27) | 19 (19)
Rash pustular (Infections and infestations) | 25 (26) | 16 (16)
Skin candida (Infections and infestations) | 14 (14) | 11 (11)
Otitis media acute (Infections and infestations) | 6 (6) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 281 (317) | 132 (139)
Vomiting (Gastrointestinal disorders) | 25 (25) | 13 (13)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 36 (37) | 28 (31)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 37 (37) | 16 (17)
Rash papular (Skin and subcutaneous tissue disorders) | 20 (22) | 11 (13)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 17 (18) | 7 (7)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 12 (12) | 11 (11)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 17 (17) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 95 (103) | 39 (39)
Pyrexia (General disorders) | 31 (31) | 16 (16)
Thermal burn (Injury, poisoning and procedural complications) | 9 (9) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT03197376/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/76/NCT03197376/SAP_001.pdf